## **Study Title** MATRIX-002: Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

Protocol Version V1.0 24May2023

NCT Number: NCT06046053

Document Date: 24May2023

## Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

MATRIX: A USAID Project to Advance the Research and Development of Innovative HIV Prevention Products for Women

Funding Agency:
US Agency for International Development (USAID)

Award/Grant Number(s):
Cooperative Agreement #7200AA22CA00002

**A Non-IND Study** 

Pharmaceutical Collaborator:
University of Pittsburgh (Pitt) / Magee-Womens Research Institute and Foundation
(MWRIF)

Protocol Co-Chair: Nyaradzo M. Mgodi, MBChB, MMed

> Protocol Co-Chair: Alexandra Minnis, PhD

> > Version 1.0

24 May 2023







# Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

## **TABLE OF CONTENTS**

| LI | ST OF A | ABBREVIATIONS AND ACRONYMS | . v |
|----|------------|------------------------------------------------|-----|
| | | DL TEAM ROSTER | |
| ΙN | VESTIC | GATOR SIGNATURE FORM | ιvi |
| PF | ROTOCO | DL SUMMARYx | vii |
| 1 | | KEY ROLES | |
| | 1.1 | Protocol Identification | |
| | 1.2 | Funding Agency and Monitor Identification | |
| | 1.3 | Laboratory(ies) | |
| | 1.4 | Data Management | |
| | 1.5 | Clinical Research Management | |
| 2 | | INTRODUCTION | |
| | 2.1 | Background | |
| | 2.2 | Description of Placebo Prototype Vaginal Films | |
| | 2.3 | Acceptability of Vaginal Film Formulations | |
| | 2.4 | Rationale for Study Design | |
| 3 | | OBJECTIVES | |
| | 3.1 | Primary Objective | |
| | 3.2 | Secondary Objectives | |
| | 3.3 | Exploratory Objectives | |
| 4 | | STUDY DESIGN | |
| | 4.1 | Identification of Study Design | |
| | 4.2 | Summary of Major Endpoints | |
| | 4.3 | Description of Study Population | |
| | 4.4 | Time to Complete Accrual | |
| | 4.5 | Study Groups | |
| | 4.6 | Expected Duration of Participation | |
| _ | 4.7 | Sites | |
| 5 | | STUDY POPULATION | |
| | 5.1 | Selection of the Study Population | |
| | 5.2 | Inclusion Criteria | |
| | 5.3 | Exclusion Criteria | |
| _ | 5.4 | Co-enrollment Guidelines | |
| 6 | 6.1 | STUDY PRODUCT | |
| | - | Regimen | |
| | 6.2 | Administration | |
| | 6.3 | Study Product Formulation and Storage | |
| | 6.4<br>6.5 | Supply and Accountability | |
| | | Ancillary Study Supplies | |
| | 6.6 | Concomitant Medications | |
| | 6.7 | Prohibited Medications, Products and Practices | тЗ |

| 7 | | STUDY PROCEDURES | 14 |
|---|---|---|---|
| | 7.1 | Screening Visit | 14 |
| | 7.2 | Enrollment Visit – Visit 2 (Day 0) | 15 |
| | 7.3 | Follow-up Visits/Contacts | |
| | 7.4 | Follow-up Procedures for Participants Who Permanently Discontinue Study Product. | 22 |
| | 7.5 | Interim Visits/Contacts | |
| | 7.6 | Behavioral Evaluations | |
| | 7.7 | Protocol Adherence Counseling | |
| | 7.8 | Clinical Evaluations and Procedures | |
| | 7.9 | Laboratory Evaluations | |
| | 7.10 | Specimen Management | |
| | 7.11 | Laboratory Oversight | |
| | 7.12 | Biohazard Containment | |
| 8 | , | ASSESSMENT OF SAFETY | |
| Ŭ | 8.1 | Safety Monitoring | |
| | 8.2 | Clinical Data and Safety Review | |
| | 8.3 | Adverse Events Definitions and Reporting Requirements | |
| | 8.4 | Pregnancy and Infant Outcomes | |
| | 8.5 | Regulatory Requirements | |
| | 8.6 | Social Harms Reporting | |
| 9 | 0.0 | CLINICAL MANAGEMENT | |
| 9 | 9.1 | Grading System | _ |
| | 9.2 | Dose Modification Instructions | |
| | 9.3 | General Criteria for Permanent Discontinuation of Study Product | |
| | 9.4 | Permanent Discontinuation in Response to Observed Adverse Events | |
| | 9.5 | Other Clinical Findings | |
| | 9.5 | HIV Infection | |
| | 9.0 | Pregnancy | |
| | - | | |
| 10 | 9.8 | Criteria for Early Termination of Study Participation | |
| 10 | | | |
| | 10.1 | Overview and Summary of Design | 34 |
| | 10.2 | Study Endpoints | |
| | 10.3 | Sample Size and Power Calculations | |
| | 10.4 | Randomization Procedures | |
| | 10.5 | Participant Accrual, Follow-up and Retention | |
| | 10.6 | Data and Safety Monitoring and Analysis | |
| 11 | _ | DATA HANDLING AND RECORDKEEPING | |
| | 11.1 | Data Management Responsibilities | |
| | 11.2 | Source Documents and Access to Source Data/Documents | |
| | 11.3 | Quality Control and Quality Assurance | |
| 12 | | CLINICAL SITE MONITORING | |
| 13 | | HUMAN SUBJECTS PROTECTIONS | |
| | 13.1 | Institutional Review Boards/Ethics Committees | |
| | 13.2 | Protocol Implementation | |
| | 13.3 | Study Coordination | |
| | 13.4 | Risk Benefit Statement | |
| | 13.5 | Informed Consent Process | |
| | 13.6 | Participant Confidentiality | 44 |

| 13.7 | Special Populations4 | 4 |
|---|---|---|
| 13.8 | Compensation 4 | 5 |
| 13.9 | Reporting4 | |
| | Access to HIV-related Care | |
| | Study Discontinuation4 | |
| 14 | PUBLICATION POLICY4 | 6 |
| 15 | APPENDICES4 | |
| APPENDI | X I: SCHEDULE OF STUDY VISITS AND EVALUATIONS4 | 7 |
| | X II: ALGORITHM FOR HIV TESTING – SCREENING/ENROLLING/FOLLOW-UP 4 | |
| APPENDIX | X III: SAMPLE INFORMED CONSENT FORM (SCREENING, ENROLLMENT, LONG-TERM | |
| STORAGE | E AND FUTURE TESTING)5 | 0 |
| APPENDI: | X IV: SAMPLE INFORMED CONSENT FORM (SEXUAL PARTNER SUBSET) 6 | 9 |
| | CES | |
| | LIST OF FIGURES | |
| ETGLIRE 1 | L: STUDY VISIT SCHEDULEXVII | ſΤ |
| | 2: STUDY PRODUCT REGIMEN | |
| | 3: STUDY VISIT SCHEDULE | |
| I TOOKE 5 | 7. 31051 11011 301125022 | • |
| | LIST OF TABLES | |
| TABLE 1: | SCREENING VISIT | 5 |
| | ENROLLMENT VISIT – VISIT 2 (DAY 0) | |
| TABLE 3: | PHONE CHECK-IN (24-72 HOURS AFTER 1 <sup>ST</sup> INSERTION) – VISIT 3 1 | 7 |
| TABLE | 4: 1-WEEK AND 2-WEEK TELEPHONE CONTACTS – VISITS 4 AND 5 (7 AND 14 DAYS | • |
| AFTI | ER VISIT 2) | 7 |
| | 4-WEEK VISIT – VISIT 6 (28 DAYS AFTER VISIT 2) | |
| | PHONE CHECK-IN (24-72 HOURS AFTER 2ND INSERTION) - VISIT 7 1 | |
| | 6-WEEK TELEPHONE CONTACT – VISIT 8 (14 DAYS AFTER VISIT 6) 2 | |
| | 8-WEEK VISIT – VISIT 9 (28 DAYS AFTER VISIT 6) 2 | |
| | FINAL CONTACT/SEV - VÌSIT 10 (7 DAYS AFTER VISIT 9) 2 | |
| TABLE 10 | ): IDI VISIT WITH SEXUAL PARTNER SUBSET 2 | 2 |
| TABLE 11 | L: SUMMARY OF BEHAVIORAL ASSESSMENTS2 | 4 |
| TABLE 12 | 2: RANGE OF POTENTIAL EFFECT SIZES FOR EACH ENDPOINT | 6 |

## Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### LIST OF ABBREVIATIONS AND ACRONYMS

ACRO African Clinical Research Organisation

AE Adverse event

AIDS Acquired immunodeficiency syndrome

ALT Alanine transaminase

API Active pharmaceutical ingredient AST Aspartate aminotransferase

BV Bacterial vaginosis

CAB Community advisory board CBC Complete blood count

CDC Centers for Disease Control and Prevention (US)

CDM Clinical data manager
CFR Code of Federal Regulations

CLIA Clinical Laboratory Improvement Act

CQA Critical quality attributes

CRF Case report form

CRM Clinical research manager
CRS Clinical research site
CT Chlamydia trachomatis

CV Cervicovaginal
CVF Cervicovaginal fluid
DAIDS Division of AIDS

DRA Drug regulatory authority

ECS-HSR Education and Compliance Support for Human Subject Research

FDA U.S. Food and Drug Administration

GC Neisseria gonorrhea GCP Good Clinical Practice

GDP Good Documentation Practices GMP Good Manufacturing Practice GRAS Generally regarded as safe

HHRC Harare Health and Research Consortium

HIPAA Health Insurance Portability and Accountability Act

HIV Human Immunodeficiency Virus
IATA International Air Transport Association

ICH E6 International Conference for Harmonization Guideline for Good Clinical Practice

IDI In-depth interview

IEC Independent Ethics Committee
IND Investigational New Drug
IoR Investigator of Record
IRB Institutional Review Board
ISP Independent Safety Physician

IUD Intrauterine device

KEMRI Kenya Medical Research Institute

KOH Saline/potassium hydroxide

LDMS Laboratory Data Management System

LTFU Loss-to-follow-up

MWRIF Magee-Womens Research Institute and Foundation

NAAT Nucleic acid amplification test NIH National Institutes of Health

OHRP Office for Human Research Protections

PEP Post-exposure prophylaxis PHI Protected health information

PI Principal Investigator

PID Pelvic inflammatory disease PrEP Pre-exposure prophylaxis PSRT Protocol Safety Review Team

PTID Participant identifier
QA Quality assurance
QC Quality control

RTI Reproductive tract infection SAE Serious adverse event

SEV Study Exit Visit

SMS Short message service

SOP Standard operating procedures

SSA Sub-Saharan Africa

SSP Study specific procedures STI Sexually transmitted infection

UPT Urine pregnancy test

USAID US Agency for International Development

UTI Urinary tract infection

VALUE Vaginal film as A Low-cost, User-administered, and Extended-release product

Wits RHI Wits Reproductive Health and HIV Institute

## Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### PROTOCOL TEAM ROSTER

#### **Protocol Co-Chair**

Nyaradzo M. Mgodi, MBChB, MMed Protocol Co-Chair

Zengeza Clinical Research Site (CRS) 7723 Cheuka Street Zengeza 3 Clinic Chitungwiza, Zimbabwe

Phone: +263-772-264616 Email: nmgodi@uz-ctrc.org

#### **Protocol Co-Chair**

Alexandra Minnis, PhD Protocol Co-Chair

RTI International 2150 Shattuck Avenue, Suite 800 Berkeley, CA 94704 USA

Phone: 1-919-485-1323 Email: aminnis@rti.org

### **Clinical Research Site (CRS) Investigators**

## University of Pittsburgh (Pitt)/Magee-Womens Research Institute and Foundation (MWRIF) CRS

## Katherine Bunge, MD, MPH Site Investigator of Record

Department of Obstetrics, Gynecology and Reproductive Sciences University of Pittsburgh School of Medicine 300 Halket Street

Pittsburgh, PA 15213 USA Phone: 412-641-6967 Fax: 412-641-1133

Email: kbunge@mail.magee.edu

## Ingrid Macio, PA-C Site Investigator

Department of Obstetrics, Gynecology and Reproductive Sciences University of Pittsburgh School of Medicine 300 Halket Street Pittsburgh, PA 15213 USA

Phone: 412-641-4242
Fax: 412-641-2319
Email: maciis@upmc.edu

#### Harare Health and Research Consortium (HHRC) CRS

## Nyaradzo M. Mgodi, MBChB, MMed Site Investigator of Record

Zengeza CRS 7723 Cheuka Street Zengeza 3 Clinic Chitungwiza, Zimbabwe Phone: +263-772-26461

Phone: +263-772-264616 Email: nmgodi@uz-ctrc.org

#### The Aurum Institute CRS

## Raesibe Agnes Pearl Selepe, MBChB Site Investigator of Record

Klerksdorp Clinical Research Centre 201 Jade Square Centre Cnr Margaretha Prinsloo and OR Tambo Drive Klerksdorp, North West Province South Africa 2571

Phone: +27 87 135 1596 Fax: +27 87 231 4977

Email: pselepe@auruminstitute.org

## Heeran Makkan, MSc Site Investigator

Tembisa CRS
Corner Rev RTJ Namane and Flint Mazibuko Drive
Tembisa Hospital, Hospital View, Tembisa
Johannesburg, Gauteng
South Africa 1632

Phone: +27 10 590 1331

Email: hmakkan@auruminstitute.org

## Wits Reproductive Health and HIV Institute (Wits RHI) CRS

## Thesla Palanee-Phillips, MMedSci, PhD, MSc Site Investigator

Wits RHI Research Centre 7 Esselen Street, 3<sup>rd</sup>-5<sup>th</sup> Floors Hillbrow, Johannesburg South Africa 2038 Phone: +2711 358 5471

Fax: +2711 336 3471 Fax: +2786 554 1093 Email: tpalanee@wrhi.ac.za

## Nkosiphile Ndlovu, MBChB, HIV Dip Man (SA) Site Investigator of Record

Wits RHI Research Centre 7 Esselen Street, 3<sup>rd</sup>-5<sup>th</sup> Floors Hillbrow, Johannesburg South Africa 2038

Phone: +2784 722 5877 Email: nkndlovu@wrhi.ac.za

## Kenya Medical Research Institute (KEMRI) CRS

## Kenneth Ngure, PhD Site Investigator

Jomo Kenyatta University of Agriculture and Technology (JKUAT)-College of Health Sciences P.O. Box 19704-00202

Nairobi, Kenya

Phone: 254-722362219 Email: Kngure@pipsthika.org

## Nelly Rwamba Mugo, MBChB, MMed, MPH Site Investigator of Record

Kenya Medical Research Institute (KEMRI) OAU Road Thika, Kenya

Phone: 254-733629665 Email: rwamba@uw.edu

#### **Sharon Hillier, PhD**

### **MATRIX Executive Director and Clinical Trials Hub Co-lead**

Magee-Women's Research Institute and Foundation (MWRIF)

204 Craft Avenue, Room B511 Pittsburgh, PA 15213 USA Phone: 1-412-641-6435

Fax: 1-412-641-6170

Email: hillsl@mwri.magee.edu

## Thesla Palanee-Phillips, PhD, MSc MATRIX Deputy Director

Wits Reproductive Health and HIV Institute (Wits RHI) Hillbrow Health Precinct

22 Esselen Street

Johannesburg, 2001 South Africa

Phone: 27-11-358-5471 Fax: 27-086-554-1093 Email: tpalanee@whri.ac.za

## Nyaradzo M. Mgodi, MBChB, MMed MATRIX Clinical Trials Hub Co-lead

Harare Health and Research Consortium (HHRC)

4 Ascot Road, Avondale

Harare, Zimbabwe

Phone: 263-24-2704920 Fax: 263-24-2704897 Email: nmgodi@uz-ctrc.org

## Leila E. Mansoor, B.Pharm, PhD MATRIX Design to Delivery (D2D) Pillar 2 Co-lead

Centre for the AIDS Programme of Research in South Africa (CAPRISA) University of KwaZulu-Natal, 2<sup>nd</sup> Floor, Doris Duke Medical Research Institute 719 Umbilo Road

Durban, KwaZulu-Natal, 4001 South Africa

Phone: 27-(0)31-655-0517

Email: Leila.Mansoor@caprisa.org

### Alexandra Minnis, PhD MATRIX D2D Pillar 2 Co-lead

RTI International 2150 Shattuck Avenue, Suite 800 Berkeley, CA 94704 USA

Phone: 1-919-485-1323 Email: aminnis@rti.org

## Catherine Chappell, MD Protocol Safety Physician

Department of Obstetrics, Gynecology and Reproductive Sciences

University of Pittsburgh 300 Halket Street Pittsburgh, PA 15213

Phone: 412-641-1403

Email: chappellca@upmc.edu

## Leslie Meyn, PhD Biostatistician/Epidemiologist

**MWRIF** 

204 Craft Avenue Pittsburgh, PA 15213 Phone: 412-641-4233 Fax: 412-641-1133

Email: meynla@mwri.magee.edu

## Tracy Zamborsky Data Manager

**MWRIF** 

204 Craft Avenue

Pittsburgh, Pennsylvania 15213 USA

Email: zambtx@upmc.edu

## Edward Livant, BSMT (ASCP), MPH MATRIX Laboratory Quality Assurance/Quality Control (QA/QC) Coordinator

**MWRIF** 

204 Craft Avenue, Room A536 Pittsburgh, PA 15213 USA Phone: 412-641-3772

Fax: 412-641-5290

Email: elivant@mwri.magee.edu

## May Beamer, BS Laboratory Manager/Supervisor

**MWRIF** 

204 Craft Avenue

Pittsburgh, PA 15213 USA

Phone: 412-641-6042 Fax: 412-641-6170

Email: mbeamer@mwri.magee.edu

## Ingrid Macio, PA-C MATRIX Clinical Research Manager (CRM)

**MWRIF** 

204 Craft Avenue Pittsburgh, PA 15213 USA Phone: 412-641-5455

Fax: 412-641-2319 Email: maciis@upmc.edu

## Sharon Riddler, MD, MPH Independent Safety Physician (ISP)

Division of Infectious Diseases University of Pittsburgh School of Medicine Keystone Building, Suite 510 3520 Fifth Avenue Pittsburgh, PA 15213 USA

Phone: 412-383-1741 or 412-383-1675

Fax: 412-383-2900 Email: riddler@pitt.edu

#### **USAID**

## Shannon Allen, PhD MATRIX Agreement Officer Representative (AOR)

Bureau of Global Health, Office of HIV AIDS, Research Division, USAID 500 D Street Southwest Washington, DC 20547 USA

Phone: 1-202-916-2201 Email: shallen@usaid.gov

## Mary Latka, PhD, MPH Chief, Microbicides Branch

Bureau of Global Health, Office of HIV AIDS, Research Division, USAID 500 D Street Southwest Washington, DC 20547 USA Email: mlatka@usaid.gov

## Kristin Vahle, MPH Project Program Analyst

Bureau of Global Health, Office of HIV AIDS, Research Division, USAID 500 D Street Southwest Washington, DC 20547 USA Email: kvahle@usaid.gov

### Pitt / MWRIF

#### Lisa C. Rohan, PhD

## VALUE (Vaginal film as A Low-cost, User-administered, and Extended-release product) Project Principal Investigator (PI)

Department of Pharmaceutical Sciences University of Pittsburgh School of Pharmacy Magee-Womens Research Institute 204 Craft Avenue Pittsburgh, PA 15213 USA

Phone: 1-412-641-6108 Fax: 1-412-641-6170

Email: Irohan@mwri.magee.edu

## Sravan K. Patel, PhD VALUE Project Co-PI

Department of Pharmaceutical Sciences University of Pittsburgh School of Pharmacy Magee-Womens Research Institute 204 Craft Avenue Pittsburgh, PA 15213 USA

Phone: 1-412-641-8276 Fax: 1-412-641-6170

Email: patels10@mwri.magee.edu

## Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### **INVESTIGATOR SIGNATURE FORM**

Version 1.0; 24 May 2023

MATRIX: A USAID Project to Advance the Research and Development of Innovative HIV Prevention Products for Women

#### Funded by:

US Agency for International Development (USAID)

#### A Non-IND Study

I, the Investigator of Record, agree to conduct this study in full accordance with the provisions of this protocol and all applicable protocol-related documents. I agree to conduct this study in compliance with United States (US) Health and Human Service regulations (45 CFR 46); USAID regulations (2 CFR 200 and 22 CFR 225); standards of the International Conference for Harmonization Guideline for Good Clinical Practice (ICH E6); Institutional Review Board/Independent Ethics Committee (IRB/IEC) determinations; all applicable in-country, state, and local laws and regulations; and other applicable requirements (e.g., USAID) and institutional policies.

I agree to maintain all study records in accordance with protocol-specified protections of participants' confidentiality and with site IRB/IEC policies and procedures. Study records must be maintained on-site for the entire implementation period of the study and a minimum of at least three years after completion of research. Pitt/MWRIF will inform the investigator/institution as to when these documents no longer need to be retained.

I have read and understand the information in this protocol, including the potential risks and side effects of the products under investigation, and will ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed about the obligations incurred by their contribution to the study.

| Name of Investigator of Record (print) | ) |
|----------------------------------------|------|
| Signature of Investigator of Record | Date |

## Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### PROTOCOL SUMMARY

**Short Title:** VALUE Placebo Film Study

**Pharmaceutical** 

**Collaborator:** Pitt/MWRIF

**Funders:** USAID

Protocol Co-Chair: Nyaradzo M. Mgodi, MBChB, MMed

Protocol Co-Chair: Alexandra Minnis, PhD

**Sample Size:** MATRIX-002 will enroll approximately 100 evaluable participants. MATRIX-

002 will also enroll a subset of up to 30 sexual partners of evaluable

participants for in-depth interviews (IDI).

**Study Population:** HIV seronegative adult (18-45 years old) persons assigned female sex at

birth who are at low risk of acquiring HIV infection (henceforth referred to

as "participants"), and sexual partners of evaluable participants

(henceforth referred to as "sexual partners").

**Study Sites:** Five sites in the US and sub-Saharan Africa (SSA):

University of Pittsburgh (Pitt)/Magee-Womens Research Institute and

Foundation (MWRIF) clinical research site (CRS);

Aurum Institute CRS;

Harare Health and Research Consortium (HHRC) CRS;

Wits Reproductive Health and HIV Institute (Wits RHI) CRS; and

Kenya Medical Research Institute (KEMRI) CRS.

**Study Design:** Two-arm, randomized, multi-center trial of monthly vaginal administration

of two placebo prototype films.

**Study Duration:** Approximately nine weeks of follow-up per participant is planned with a

projected accrual period of approximately 3-6 months. The total duration of

the study will be approximately 6-9 months.

**Study Products:** Placebo vaginal films A and B, 2" x 2" in size, which differ by shape.

**Study Regimen:** Participants will be randomized (1:1) to insert either placebo vaginal film A

or placebo vaginal film B once monthly for two months.

Figure 1: Study Visit Schedule



### **Primary Objective:**

### **Acceptability**

• To assess the acceptability of two placebo film types (A and B) when administered vaginally once monthly for two months.

## **Primary Endpoint:**

#### **Acceptability**

• Participant ratings of overall satisfaction with use of the placebo vaginal films.

#### **Secondary Objectives:**

#### Safety

• To assess the safety of two placebo film types (A and B) when administered vaginally once monthly for two months.

#### **Usability**

To assess participants' ability to properly insert the placebo vaginal film.

#### **Secondary Endpoints:**

#### Safety

• Proportion of participants with genitourinary Grade 2 or higher Adverse Events deemed related to study product.

### Usability

• Proportion of participants with clinically assessed proper insertion (more than half of the vaginal film proximal to introitus).

### **Exploratory Objectives:**

### Participant acceptability, attitudes and experiences

• To explore multiple dimensions of acceptability of two placebo film types (A and B) and participants' attitudes towards and experiences with the vaginal film.

## **Sexual partner attitudes and experiences**

• To explore sexual partners' attitudes towards and experiences with the vaginal film.

### **Vaginal microenvironment**

• To assess the impact of placebo film use on participants' vaginal microenvironment when administered vaginally once monthly for two months.

#### Social harms and social benefits

• To describe the reported experiences of social harms and social benefits over the course of vaginal film use.

### **Exploratory Endpoints:**

### Participant acceptability, attitudes and experiences

- Participant responses to quantitative acceptability assessments and IDI questions. Multiple dimensions will be explored, including:
  - Vaginal film attributes, including acceptability (e.g., ease of insertion, burden, perceived effectiveness of film as delivery form) and preferences
  - Experience and comfort with inserted vaginal film (e.g., expulsions, leakage, awareness of film during daily activities)
  - Experience during sex and menses
  - o Vaginal practices and concomitant vaginal product use while using vaginal film
  - o Perception of sexual partners' attitudes towards vaginal film
  - Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option
  - o Interest in using vaginal film as a future HIV prevention option

#### **Sexual partner attitudes and experiences**

- Sexual partner responses during IDI related to:
  - Vaginal film attributes, including acceptability and preferences
  - Perception of participant's experience using the vaginal film during the study
  - Physical sensation of the participant's vaginal film use during sex (as relevant)
  - Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option

#### **Vaginal microenvironment**

- Change from baseline in vaginal pH following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in quantity of selected vaginal microbiota following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in Nugent score following film use during the two study phases (i.e., with and without sexual abstinence requirement).

#### **Social harms and social benefits**

- Participant self-report of social harms (i.e., non-clinical adverse consequences of study participation or product use that may manifest in social, psychological or physical ways).
- Participant or sexual partner self-report of social benefits (e.g., positive consequences of product use disclosure, self-confidence, improved communication with intimate partner) resulting from vaginal film use and/or study participation.

#### 1 KEY ROLES

#### 1.1 Protocol Identification

Protocol Title: Trial to Assess Acceptability and Safety of Two Placebo Prototype

Vaginal Films

Protocol Number: MATRIX-002

Short Title: VALUE Placebo Film Study

Date: 24 May 2023

## 1.2 Funding Agency and Monitor Identification

Funding Agency: USAID

Bureau of Global Health, Office of HIV/AIDS, Research Division

500 D Street Southwest Washington, DC 20547 USA

Pharmaceutical Collaborator: Pitt/MWRIF

204 Craft Avenue

Pittsburgh, PA 15213 USA

Monitor – African sites: African Clinical Research Organisation (ACRO)

Phase 3, Second Floor Offices, Centurion Science Park, 1011 Pretorious Avenue, Lyttelton Manor, Centurion, 0157

South Africa

Monitor – US site: University of Pittsburgh Education and Compliance Support for

Human Subject Research (ECS-HSR)

Office of Research Protections Heiber Building, Suite 401

3500 Fifth Avenue,

Pittsburgh, PA 15213 USA

## 1.3 Laboratory(ies)

MATRIX/MWRIF 204 Craft Avenue

Pittsburgh, Pennsylvania 15213 USA

## 1.4 Data Management

Quantitative Data Center: MATRIX/MWRIF

204 Craft Avenue

Pittsburgh, Pennsylvania 15213 USA

Qualitative Data Center: RTI International

2150 Shattuck Avenue, Suite 800

Berkeley, CA 94704 USA

## 1.5 Clinical Research Management

MATRIX/MWRIF 204 Craft Avenue

Pittsburgh, Pennsylvania 15213 USA

#### 2 INTRODUCTION

## 2.1 Background

Topical microbicides are agents designed to prevent or at least substantially reduce the risk of sexual acquisition and transmission of HIV when applied to the genital or rectal mucosa. Vaginal films are an attractive dosing option for topical (vaginal) delivery of anti-HIV drugs. In terms of costs of production and manufacturing, films are relatively inexpensive, scalable, physically and chemically stable, and amenable to a range of active ingredients including combinations of excipients. In terms of use, films are discreet, portable, and easy to store. Vaginal films can deliver fixed doses of pharmacologically active agents with minimal mess or leakage and without an applicator. Due to their small volume, films also generate no significant alterations in innate microbiome as shown in previous clinical evaluation for our FAME program (U19 AI082639<sup>1</sup>, U19 AI120249<sup>2</sup>), and incur less dilution of endogenous antiviral or antibacterial properties in vaginal fluids as compared to vaginal gels. Feedback from women in several clinical and focus-group studies - NCT01231763 (FACE)<sup>3</sup>, NCT02908503 (FLAG)<sup>4</sup>, NCT02602366 (Quatro)<sup>5</sup>, PASII<sup>6</sup>, NCT01334827 (MIST)<sup>7,8</sup>, NCT01548560 (FAME 02)<sup>9</sup>, FAME 02B<sup>10</sup>, NCT02579083 (VAST)<sup>11</sup>, NCT01989663 (FAME 04)<sup>12</sup>, NCT02280109 (FAME 05)<sup>13</sup>, NCT03537092 (FAME 101)<sup>14</sup>, FAME 102 (unpublished data), NCT04319718 (FAME 103)<sup>15</sup>, NCT04391036 (FAME 103B)<sup>16</sup> – supported the willingness for women to use such products and the advancement and development of vaginal films for discrete HIV prevention. 5,6,9-11

The long-term goal of the VALUE (Vaginal film as A Low-cost, User-administered, and Extended-release product) project is to develop and evaluate an extended-release vaginal film containing dapivirine, a potent NNRTI, which could provide protection from HIV for at least one month following a single application. Previously, the Pitt/MWRIF team developed and evaluated quick dissolve films for on-demand vaginal administration of several anti-HIV drug candidates including dapivirine. Hard was also confirmed the feasibility of design of a monthly film platform (LATCH R61/33 AI142687)<sup>17</sup> in a nonhuman primate (macaque) model. Furthermore, retention of films within the vagina was established during menses and sex in the macaque model. The VALUE project aims to design a one-month vaginal film containing dapivirine as the active pharmaceutical ingredient (API) to provide a low cost and convenient option for women for protection from HIV infection through sex. Previous studies have supported the acceptability and safety of the quick dissolve and 7-day sustained release films, but there is limited data regarding a monthly vaginal film.

MATRIX-002 is a randomized trial assessing the acceptability and safety of two vaginal placebo film products that differ in shape. Specifically, the 2"x2" films differ with respect to shape of the corners. One film product is square in shape, while the second product has rounded edges on all four corners. These differences may impact product acceptability and usability. The proposed study will evaluate the acceptability, safety, and self-insertion success of these 1-month placebo film products when applied vaginally with and without sex at five clinical sites, one in the United States and four in South Africa, Zimbabwe, and Kenya. Building on the existing evidence base for the quick dissolve and 7-day extended-release films, multiple African sites will participate in MATRIX-002 alongside the US site, affording the opportunity to obtain critical information and feedback from women who have the greatest potential to benefit from access to a range of HIV prevention products. This study of the one-month placebo vaginal film will examine overall

satisfaction with the film after using it, multiple components and correlates of acceptability, as well as topics relevant to adherence and preference. The design of these assessments is informed by a recent systematic review of the Theoretical Framework of Acceptability (Sekhon), <sup>18</sup> published by Ortblad et al. <sup>19</sup>

Additionally, by investigating the attitudes and experiences that sexual partners had while MATRIX-002 participants used the vaginal film, this study hopes to gain a deeper understanding of how partners' opposition or support may affect a user's ability to safely, correctly and consistently use a vaginal film for HIV prevention in the future. This, in turn, can contribute to efforts to mitigate concerns and cultivate support among men for HIV prevention research, HIV prevention products, and microbicide use. Data from in-depth interviews (IDI) may also provide insight to the strategies and counseling messages that could be used in couples' education and counseling for future trials, with the objective of promoting use of the vaginal film.

### 2.2 Description of Placebo Prototype Vaginal Films

## 2.2.1 Placebo Vaginal Film A

Placebo Vaginal Film A is made of film-forming polymers, release-modifying polymers, and plasticizers. It differs from Placebo Vaginal Film B by the shape (square vs. rounded edges). All the excipients used have a history of pharmaceutical use (https://www.accessdata.fda.gov/scripts/cder/iig/index.cfm). The formulations contain multiple excipients, namely, hydroxypropyl cellulose, Hypromellose, hydroxyethyl cellulose, ammonio methacrylate copolymer type B, propylene glycol, and polyethylene glycol. A vaginal film containing similar excipients was utilized in the FAME 101 study (ClinicalTrials.gov Identifier: NCT03537092)<sup>14</sup> without any adverse outcomes in healthy participants.

#### 2.2.2 Placebo Vaginal Film B

Placebo Vaginal Film B is also made of film-forming polymers, release-modifying polymers, and plasticizers. It differs from Placebo Vaginal Film A by the shape (square vs. rounded edges).

#### 2.3 Acceptability of Vaginal Film Formulations

End-user acceptability of vaginal films as an option for women has been confirmed through input from nearly 3000 women. <sup>5,6,9-11</sup> Prior end-user acceptability data was collected primarily through programs evaluating HIV prevention products to gain insight regarding the acceptability of the vaginal film platform when applied for HIV prevention. Some of the data also include preferences associated with multipurpose prevention platforms. In these studies, we have obtained data comparing films with other dosage forms, explored end-user acceptability in the context of sexual intercourse and obtained information from end-users that has directed our target critical quality attributes (CQAs) including size, color and texture. We also gained insights that informed film use instructions and explored the relationship between formulation modification, end-user acceptability, and ease of use experiences with the product. Overall, women have found the vaginal film platform to be acceptable and easy to use.

### 2.4 Rationale for Study Design

The primary objective of this study is to assess the acceptability of two placebo film types (A and B) when administered vaginally once monthly for two consecutive months. Previous research has supported the safety of the film excipients, but there is little data on the acceptability of a monthly vaginal film. The study is designed to assess acceptability parameters in the first month in ideal conditions (i.e., pelvic rest). During this phase, we anticipate that participants will be unaware of the film's presence in the vagina based on prior clinical research with vaginal film products; however, it is possible that with time the film might contribute to discharge as it dissolves and/or be expelled during menses. The first month, during which participants are instructed to refrain from putting anything into the vagina, will provide valuable insight into user experiences with the film without extraneous interruptions. The second month, during which participants are allowed to have sexual intercourse and use vaginal products, will provide important information about user experience with the film with vaginal stimuli. We anticipate that the film will stay in place despite potential disruptors but can only understand this through the second month of use. By evaluating two placebo films we hope to understand if there are differences in performance (e.g., acceptability and insertion success) and what attributes potentially contribute to these outcomes. Aspects of the film that lead to better performance will be incorporated into future film design.

This study has been designed to add to our knowledge about potential end-users' acceptability of and perceptions towards long-term (1 month) use of films with different shapes. Acceptability will be assessed through quantitative questionnaires and IDIs with users and, among a subset, IDIs with their sexual partners. Instructional materials will be utilized to familiarize users with the insertion process. These materials were designed based on participant feedback from previous trials. Product misplacement such as partial insertion has been noted in clinical trials of vaginal films previously conducted at the University of Pittsburgh.<sup>4</sup> While most participants could successfully insert the vaginal films, incorrect film placement was noted for some. In some instances, the vaginal film stuck to the finger after attempted insertion and in other instances the film was visualized on the external genitalia, which illustrates the importance of assessing ease of proper insertion and film attributes relevant to usability in this placebo study. Since the film is intended to provide HIV protection for a month after a single application, identification of any adverse effects will also be an integral part of this study. Importantly, experiences of the participants and their partners in the context of sex will also be explored. Previous studies have found the vaginal film to be safe and acceptable as quick dissolve and 7-day sustained release formulations, but the 1-month long vaginal film has never been tested in women. This placebo study will provide critical information on acceptability, safety, usability, and user experience, which will be incorporated in the dapivirine film development and clinical evaluation program. Finally, although NCT02702895 (MTN-032) and other studies have shown that male partners play an important role in women's adherence to microbicides,<sup>20</sup> more research is needed to understand how this manifests specifically in the context of women's use of extended-release vaginal films. Therefore, perceptions of the vaginal film will also be elicited from sexual partners of study participants.

#### 3 OBJECTIVES

## 3.1 Primary Objective

#### **Acceptability**

• To assess the acceptability of two placebo film types (A and B) when administered vaginally once monthly for two months.

#### 3.2 Secondary Objectives

#### Safety

• To assess the safety of two placebo film types (A and B) when administered vaginally once monthly for two months.

#### **Usability**

• To assess participants' ability to properly insert the placebo vaginal film.

#### 3.3 Exploratory Objectives

#### Participant acceptability, attitudes and experiences

• To explore multiple dimensions of acceptability of two placebo film types (A and B) and participants' attitudes towards and experiences with the vaginal film.

### **Sexual partner attitudes and experiences**

• To explore sexual partners' attitudes towards and experiences with the vaginal film.

#### **Vaginal microenvironment**

• To assess the impact of placebo film use on participants' vaginal microenvironment when administered vaginally once monthly for two months.

#### Social harms and social benefits

• To describe the reported experiences of social harms and social benefits over the course of vaginal film use.

#### 4 STUDY DESIGN

#### 4.1 Identification of Study Design

MATRIX-002 is a two-arm, randomized, multi-center trial to assess acceptability, safety and usability of two placebo prototype films when administered vaginally once monthly for two months.

### 4.2 Summary of Major Endpoints

### **Primary Endpoints:**

#### Acceptability

• Participant ratings of overall satisfaction with using the placebo vaginal films.

#### **Secondary Endpoints:**

#### Safety

• Proportion of participants with genitourinary Grade 2 or higher Adverse Events deemed related to study product.

#### Usability

• Proportion of participants with clinically assessed proper insertion (more than half of the vaginal film proximal to introitus).

## **Exploratory Endpoints:**

#### Participant acceptability, attitudes and experiences

- Participant responses to quantitative acceptability assessments and IDI questions. Multiple dimensions will be explored, including:
  - Vaginal film attributes, including acceptability (e.g., ease of insertion, burden, perceived effectiveness of film as delivery form) and preferences
  - Experience and comfort with inserted vaginal film (e.g., expulsions, leakage, awareness of film during daily activities)
  - Experience during sex and menses
  - Vaginal practices and concomitant vaginal product use while using vaginal film
  - o Perception of sexual partners' attitudes towards vaginal film
  - Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option
  - o Interest in using vaginal film as a future HIV prevention option

#### **Sexual partner attitudes and experiences**

- Sexual partner responses during IDI related to:
  - Vaginal film attributes, including acceptability and preferences
  - o Perception of participant's experience using the vaginal film during the study
  - o Physical sensation of the participant's vaginal film use during sex (as relevant)
  - Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option

#### **Vaginal microenvironment**

- Change from baseline in vaginal pH following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in quantity of selected vaginal microbiota following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in Nugent score following film use during the two study phases (i.e., with and without sexual abstinence requirement).

#### Social harms and social benefits

- Participant self-report of social harms (i.e., non-clinical adverse consequences of study participation or product use that may manifest in social, psychological or physical ways).
- Participant and sexual partner self-report of social benefits (e.g., positive consequences of product use disclosure, self-confidence, improved communication with intimate partner) resulting from vaginal film use and/or study participation.

## 4.3 Description of Study Population

The study population will consist of HIV seronegative adult (18-45 years old) persons assigned female sex at birth who meet the criteria outlined in Sections 5.2.1 and 5.3, and sexual partners who meet eligibility criteria as described in Section 5.2.2.

#### 4.4 Time to Complete Accrual

The time to complete accrual at all sites is anticipated to be approximately 3-6 months.

#### 4.5 Study Groups

MATRIX-002 will enroll approximately 100 evaluable participants, randomized (1:1) to either placebo vaginal film A or B. MATRIX-002 will also enroll a subset of up to 30 sexual partners for an IDI. See Section 10.3 for more details.

#### 4.6 Expected Duration of Participation

Once randomized to placebo film A or B, participants will complete approximately nine weeks of follow-up. The total duration of the study will be approximately 6-9 months.

#### 4.7 Sites

The following five sites in the United States and sub-Saharan Africa (SSA) will take part in MATRIX-002: University of Pittsburgh (Pitt)/Magee-Womens Research Institute and Foundation (MWRIF) clinical research site (CRS), Aurum Institute CRS, Harare Health and Research Consortium (HHRC) CRS, Wits Reproductive Health and HIV Institute (Wits RHI) CRS, and Kenya Medical Research Institute (KEMRI) CRS.

#### 5 STUDY POPULATION

#### **5.1** Selection of the Study Population

The inclusion and exclusion criteria in Sections 5.2 and 5.3 will be used to ensure the appropriate selection of study participants. In addition, a sample of up to 30 sexual partners for whom participants have given permission to contact will be selected for participation in an IDI.

#### 5.1.1 Recruitment

Participants will be recruited from a variety of sources across sites including, but not limited to, existing databases (as permitted by local guidelines on protected health information [PHI]), primary care health clinics, family planning clinics, HIV testing facilities, gynecology clinics, institutions of higher learning, other community-based organizations, and through community outreach activities. Recruitment materials will be approved by site Institutional Review Boards/Independent Ethics Committees (IRB/IEC) prior to use per local requirements. Community education strategies, including group sessions, may be employed as part of participant/partner outreach. Sites will develop and implement local standard operating procedures (SOP) to target potential participants for recruitment.

#### 5.1.2 Retention

Once a participant is enrolled in MATRIX-002, study sites will make every effort to retain the participant in follow-up to minimize possible bias associated with loss-to-follow-up (LTFU). An average retention rate of 95% will be targeted across sites. Sites will develop and implement local SOPs to target and ensure high rates of retention.

#### 5.2 Inclusion Criteria

### **5.2.1 Participants**

Potential participants must meet all the following criteria prior to Enrollment (unless otherwise specified):

- 1) Aged 18 to 45 years (inclusive) at Screening, verified per site SOP.
- 2) Assigned female sex at birth.
- 3) Able and willing to provide written informed consent to be screened for and enrolled in MATRIX-002 in one of the study languages (as specified in site SOP).
- 4) Able and willing to provide adequate contact/locator information, as defined in site SOP.
- 5) Able and willing to comply with all protocol requirements, including:
  - Abstaining from all receptive sexual intercourse (vaginal, anal, digital, oral) for the first month of product use.
  - Abstaining from using other intravaginal products for the first month of product use.
  - Abstaining from engaging in intravaginal practices for the first month of product use.
  - Refraining from participation in other research studies for the duration of the study unless approved by the Protocol Safety Review Team (PSRT).
  - Responding to scheduled phone/short message service (SMS) contacts.
  - Attending all clinic follow-up visits.
- 6) HIV-uninfected based on testing performed at Screening and Enrollment (per protocol algorithms in Appendix II).
- 7) Per participant report, if in a relationship, must be in a mutually monogamous relationship with a partner who is not known to be HIV positive or to currently have a sexually transmitted infection (STI).

- 8) Negative urine pregnancy test at Screening and Enrollment.
- 9) Participants over the age of 21 (inclusive) must have documentation of a Grade 0 Pap smear within the past 3 years prior to Enrollment, or a Grade 1 Pap smear at Screening with no treatment required, per the Female Genital Grading Table for Use in Microbicide Studies Addendum 1 (Dated November 2007) to the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
- 10) Protected from pregnancy starting two weeks before Screening and continuing for the duration of study participation by an effective contraceptive method as confirmed by site SOP; effective methods include:
  - Hormonal methods except vaginal rings
  - Copper intrauterine device (IUD)
  - Sterilization of participant
  - Correct and consistent condom use (for US site only)
  - Abstinence from penile-vaginal intercourse

#### **5.2.2 Sexual Partners**

Potential participants for the sexual partner IDI subset must meet all of the following criteria to be eligible for inclusion in the study:

- 1. Identifies as a sexual partner of a MATRIX-002 participant.
- 2. Identified by participant as a sexual partner during MATRIX-002 for whom the participant has given permission to contact (as specified in site SOP).
- 3. Able and willing to provide written informed consent in one of the study languages (as specified in site SOP).
- 4. Able and willing to complete the required study procedures.
- 5. Must be 18 years old or above at the time of their study participation, verified per site SOP.

#### 5.3 Exclusion Criteria

Potential participants must not meet any of the following criteria prior to Enrollment (unless otherwise specified):

- 1) Per participant report at Screening and Enrollment, intends to do any of the following during the study participation period:
  - Become pregnant.
  - Breastfeed.
  - Relocate away from the study site.
  - Travel away from the study site for a time period that would interfere with product resupply and/or study participation.
- 2) Positive HIV test at Screening or Enrollment.
- 3) Positive test for *Trichomonas vaginalis* (TV), *Neisseria gonorrhea* (GC), *Chlamydia trachomatis* (CT), or *Treponema pallidum* (Syphilis) at Screening or (per participant report) treated for potential STI within past 12 months.
- 4) Diagnosed with urinary tract infection (UTI), pelvic inflammatory disease (PID), or reproductive tract infection (RTI) requiring treatment per WHO guidelines at Enrollment.

Note: Otherwise eligible participants diagnosed during screening with a UTI, symptomatic yeast infection or symptomatic BV infection are offered treatment consistent with WHO recommendations. If treatment is completed and symptoms have resolved within 45 days of obtaining informed consent for screening, the participant may be enrolled.

5) Clinically apparent Grade 2 or higher pelvic exam finding per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]) at Enrollment.

Note: Otherwise eligible participants with exclusionary pelvic exam findings at Screening may be enrolled/randomized if treatment is begun at least 7 days prior to enrollment and findings have improved to a non-exclusionary severity grading or resolved by the time of enrollment. Spotting/bleeding will be considered exclusionary only if greater than what would be expected from contraceptive use.

- 6) Participant report and/or clinical evidence of any of the following:
  - Known adverse reaction to any of the study product materials (ever).
  - Hysterectomy.
  - Surgical procedure involving the pelvis in the 30 days prior to Enrollment.
  - Use of diaphragm, NuvaRing, or (for African sites only) spermicide for contraception in the two weeks prior to Screening.
  - Antibiotic or antifungal (oral or intravaginal) therapy within 7 days of Enrollment.
  - Prior use of post-exposure prophylaxis (PEP) or oral pre-exposure prophylaxis (PrEP) (including FTC/TDF) in the 4 weeks prior to Screening or any prior use of long-acting systemic PrEP (including cabotegravir or islatravir).
  - Use of any of the following in the 12 months prior to Screening: stimulants (cocaine [including crack], methamphetamine, or non-physician prescribed pharmaceutical-grade stimulants), or inhaled nitrates, or illicit injection drug use of any kind.
  - At Screening or Enrollment, as determined by the Investigator of Record (IoR)/designee, has any significant uncontrolled active or chronic cardiovascular, renal, liver, hematologic, neurologic, gastrointestinal, psychiatric, endocrine, respiratory, immunologic disorder or infectious disease.
- 7) Has any of the following laboratory abnormalities at Screening:
  - Grade 2 or higher Aspartate aminotransferase (AST), alanine transaminase (ALT), creatinine, or Hemoglobin per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017.
- 8) Has any other condition that, in the opinion of the IoR/designee, would preclude informed consent, make study participation unsafe, complicate interpretation of study outcome data, or otherwise interfere with achieving the study objectives.

### 5.4 Co-enrollment Guidelines

Participants must not take part in other research studies involving drugs, medical devices, vaginal products, or vaccines starting two weeks before the Screening Visit and while taking part in MATRIX-002, unless approved by the PSRT. Participants must not take part in observational or qualitative studies while taking part in MATRIX-002, unless approved by the PSRT. Each site will be responsible for defining procedures for management and prevention of co-enrollment prior to initiation.

Should any participant report concurrent participation in contraindicated studies after enrolling in MATRIX-002, the IoR/designee will consult the PSRT regarding ongoing product use and other potential safety considerations associated with co-enrollment, or regarding potential product acceptability considerations associated with co-enrollment.

#### **6** STUDY PRODUCT

#### 6.1 Regimen

The products being used in this study are the placebo prototype vaginal films A and B. The two films differ by the shape (square vs. rounded edges). At each of the study sites, participants will be randomized (1:1) to receive either placebo vaginal film A or B. Each participant will receive one dose per month for two consecutive months, for a total of 2 doses of placebo vaginal film.

Figure 2: Study Product Regimen

45 days No sex or vaginal product use permitted No restrictions on sex or vaginal product permitted No restrictions on sex or vaginal permitted No restrictions or vaginal permitted No rest



#### 6.2 Administration

After eligibility is confirmed and the participant is randomized to one of two films (Placebo Film A or B) site staff will retrieve the assigned film from the pharmacy. Participants will self-insert the film at the study clinic, and film placement will be checked visually by a study clinician. If less than half of the vaginal film is proximal to introitus, participants will have the film removed and asked to try again with a new film. If less than half of the vaginal film is proximal to introitus a second time, participants will have the film removed and a third film inserted by the clinician using a speculum.

#### 6.3 Study Product Formulation and Storage

Films are composed of film-forming polymers, release modifying polymers, and plasticizers. The 2"x2" films will be packaged into foil-lined pouches and stored at room temperature. Good

Manufacturing Practice (GMP) stability testing will be conducted for the clinical trial product material as per ICH guidelines.

#### 6.4 Supply and Accountability

#### **6.4.1 Study Product Supply**

Study product will be manufactured and packaged by Benefit Coatings, Stratford, CT, in compliance with cGMP. Product release testing includes GMP Microbial Limits Testing (USP61/62). After product release, the packaged study product will be provided to the clinical sites.

## **6.4.2 Study Product Dispensing**

Study product will be dispensed to clinic staff only upon receipt of a written prescription signed by an authorized prescriber.

## **6.4.3 Study Product Accountability**

The clinical study site pharmacist(s) will maintain complete accountability records of all study products received for this protocol and dispensed to participants. Additional documentation will be required for study product returns, destruction (if applicable).

#### **6.4.4 Retrieval of Unused Study Products**

All unused study products must be accounted for by the site Pharmacy after the study is completed or terminated.

#### 6.5 Ancillary Study Supplies

Clinic staff will offer male condoms to all participants after the first month of vaginal film use.

#### 6.6 Concomitant Medications

All concomitant medications will be recorded on case report forms (CRF) for participants starting at Screening. Concomitant medications include any prescription, over the counter or herbal/traditional medication or preparation. Enrolled study participants may use concomitant medications during study participation but will be asked to abstain from medications and products noted as prohibited in Section 6.7.

#### **6.7 Prohibited Medications, Products and Practices**

Participants will be instructed to practice "pelvic rest" during the first month of participation. This means nothing should enter the vagina: fingers, penis, tampon, toys, etc. Participants will be asked to abstain from any penetrative sex (i.e., penile or with the use of an instrument that penetrates past the labia majora), intravaginal practices (e.g., douching), and use of all intravaginal medications and products during the first month of participation. If a participant reports receptive sexual activity, douching, or use of an intravaginal medication or product, the site staff will counsel the participant about the importance of adhering to the protocol (if reported

during first month of product use) and record these behaviors on the appropriate CRF. During the second month of participation there are no restrictions on sexual activity, intravaginal practices or products. Please reference the MATRIX-002 Study Specific Procedures (SSP) Manual for additional details.

#### 7 STUDY PROCEDURES

An overview of the study visits and evaluations schedule is provided in Appendix I. Presented in this section is additional information on visit-specific study procedures. Detailed instructions to guide and standardize procedures across sites as well as to specify the visit windows are provided in the MATRIX-002 SSP Manual.

Figure 3: Study Visit Schedule



#### 7.1 Screening Visit

Potential participants will provide written informed consent prior to any study procedures including all screening assessments to determine their eligibility to take part in the study. Participants will be counselled to abstain from sex and from use of intravaginal products (see Section 6.7) for the first month of study product use. Eligibility determination will include baseline demographics and medical history, physical and pelvic examination, urine pregnancy test (UPT), and HIV/STI screening. If eligible, potential participants will return within 45 days for their Enrollment Visit. For women with a regular menstrual cycle, the Enrollment Visit (and subsequent clinic visits if enrolled) will ideally be scheduled when the potential participant is not on her period.

Note: Multiple visits may be conducted within the screening window to complete all required screening procedures, including any procedures that need to be repeated (e.g., blood draw), if necessary.

Note: Potential participants who fail their first screening attempt may be re-screened once.

**Table 1: Screening Visit** 

| Screening Visit – Visit 1 | | |
|---|---|---|
| Component | | Procedures |
| Administrative and Regulatory Behavioral/Counseling | | <ul> <li>Obtain written informed consent for screening and enrollment (sites<br/>may split screening and enrollment consent if requested/required by<br/>IRB/IEC)</li> </ul> |
| | | Assign a unique Participant Identification (PTID) number |
| | | Assess eligibility |
| | | Collect demographic information |
| | | Collect locator information |
| | | Provide reimbursement |
| | | Schedule next visit/contact* |
| | | HIV pre- and post-test counseling |
| | | HIV/STI risk reduction counseling |
| | | Protocol counseling (including regarding pelvic rest in Month 1) |
| | | Collect medical and menstrual history |
| | | Collect concomitant medications |
| Clinical | | Perform full physical examination |
| Omnour | | Perform pelvic examination (including bimanual exam) |
| | | Treat or prescribe treatment for RTI/UTI/STIs* |
| | | Provide available test results |
| | Saliva | HIV test(s) (only at sites with CLIA certification) |
| | Urine | Urine pregnancy test |
| | | Urine dipstick/culture* |
| Laboratory | | HIV test(s) (not required for sites that conduct saliva testing) |
| | Blood | Complete blood count (CBC) |
| | | Serum creatinine |
| | | AST/ALT |
| | | Syphilis serology |
| | Pelvic | Nucleic acid amplification test (NAAT) for GC/CT/TV |
| | | Pap test^ |
| | | <ul> <li>Saline/potassium hydroxide (KOH) wet mount for candidiasis and/or<br/>bacterial vaginosis (BV)*</li> </ul> |

<sup>\*</sup>If indicated and/or per local standard of care; ^ if indicated (if participant is unable to provide documentation of a normal Pap test within 3 years prior to enrollment)

### 7.2 Enrollment Visit – Visit 2 (Day 0)

Within 45 days of the Screening Visit, willing and eligible participants will have their eligibility confirmed and be randomized (1:1) to placebo vaginal film A or B. Participants will again be counselled to abstain from sex and from use of vaginal products (see Section 6.7) for the first month of study product use. Study staff will review instructional materials about the film and film insertion with participants prior to insertion of the first film. Participants will be asked to provide a urine sample for a UPT, undergo HIV/STI screening and a pelvic examination, provide a blood sample for plasma archive, and complete an interviewer-administered baseline acceptability questionnaire about the film. Participants will then be asked to insert the film at the study clinic, and film placement will be checked visually by a study clinician. If less than half of the vaginal film is proximal to introitus, participants will have the film removed and asked to try again with a
new film. If less than half of the vaginal film is proximal to introitus a second time, participants will have the film removed and a third film inserted by the clinician using a speculum. Participant attempts to insert the film will be documented on the appropriate CRF.

Table 2: Enrollment Visit – Visit 2 (Day 0)

| | sit – Visit 2 (Day 0) | |
|---|---|---|
| Component | | Procedures |
| Administrative and Regulatory | | <ul> <li>Review informed consent or (for sites that use separate screening and<br/>enrollment consent forms if requested/required by IRB/IEC) obtain<br/>written informed consent for enrollment</li> </ul> |
| | | Assess and confirm eligibility |
| | | Review/update locator information |
| | | Randomization |
| | | Provide reimbursement |
| | | Schedule next visit/contact* |
| | | HIV pre- and post-test counseling |
| | | HIV/STI risk reduction counseling |
| Behavioral/Co | nuncalina | Protocol counseling (including regarding pelvic rest in month 1 and product use) |
| Bellavioral/OC | Juliselling | Review instructional materials |
| | | Baseline behavioral questionnaire (acceptability and risk/protective behaviors) |
| | | Post-insertion behavioral assessment |
| | | Review/update medical and menstrual history |
| | | Review/update concomitant medications |
| | | Perform targeted physical examination* |
| | | Perform pelvic examination with speculum |
| Clinical | | AE assessment |
| | | Treat or prescribe treatment for RTI/UTI/STIs* |
| | | Visual examination by clinician to check vaginal film placement |
| | | Clinician film insertion assessment |
| | 1 | Provide available test results |
| | Saliva | HIV test(s) (only at sites with CLIA certification) |
| | Urine | Urine pregnancy test |
| | Jille | Urine dipstick/culture* |
| | | HIV test(s) (not required for sites that conduct saliva testing) |
| Laboratory | | Plasma for archive |
| | Blood | • CBC* |
| | | Serum creatinine* |
| | | AST/ALT* |
| | Pelvic | NAAT for GC/CT/TV |
| | | Saline/KOH wet mount for candidiasis and/or BV* |
| | | Vaginal Gram stain |
| | | Vaginal swab(s) for microbiota |
| | | Vaginal pH |

| Enrollment Visit - Visit 2 (Day 0) | |
|---|---|
| Component | Procedures |
| Study Product/Supplies | <ul> <li>Provide vaginal film for self-insertion at clinic</li> <li>Clinician insertion of vaginal film at clinic (only if participant fails two attempts)</li> </ul> |

<sup>\*</sup>If indicated and/or per local standard of care

## 7.3 Follow-up Visits/Contacts

## 7.3.1 Phone check-in (24-72 hours after 1<sup>st</sup> insertion) – Visit 3

Between 24 and 72 hours after the insertion of the first film, a member of the study team will contact the study participant via telephone or short message service (SMS) to assess experiences with the first vaginal film *in situ*. Participants who prefer to complete these procedures in-person may elect to do so. The staff member will ask the participant about initial experiences with the film in place, any concerns about product placement and leakage, and elicit any questions or other concerns. If conducted as a phone conversation, this is anticipated to be less than 5 minutes. If conducted as an SMS exchange, this is anticipated to be less than 5 text messages from each party. If participants raise any concerns that require more in-depth discussion, the staff member will assess the proper follow-up method.

Table 3: Phone check-in (24-72 hours after 1st insertion) – Visit 3

| Phone check-in (24-72 hours after 1st insertion) – Visit 3 | |
|---|---|
| Component | Procedures |
| Administrative and Regulatory | Provide reimbursement |
| Behavioral/Counseling | Brief behavioral assessment (concerns and comfort with film use) |

## 7.3.2 1-week and 2-week Telephone Contacts – Visits 4 and 5 (7 and 14 days after Visit 2)

Approximately one week and two weeks after Enrollment, the study team will contact the study participant via telephone or SMS to assess participant wellness, comfort with the film, and any concerns. Participants who prefer to complete these procedures in-person may elect to do so. Participants who report AEs or otherwise express concerns may be asked to come in for an Interim Visit, if willing, to conduct additional counseling and/or testing as needed.

Table 4: 1-week and 2-week Telephone Contacts – Visits 4 and 5 (7 and 14 days after Visit 2)

| 1-week and 2-week Telephone Contacts – Visits 4 and 5 (7 and 14 days after Visit 2) | |
|---|---|
| Component | Procedures |
| | Review/update locator information |
| Administrative and Regulatory | Provide reimbursement |
| | Schedule next visit/contact |
| Behavioral/Counseling | Brief behavioral assessment (concerns and comfort with film use) |
| | Protocol counseling* |

| 1-week and 2-week Telephone Contacts – Visits 4 and 5 (7 and 14 days after Visit 2) | |
|---|---|
| Component | Procedures |
| | Review/update medical and menstrual history |
| Clinical | Review/update concomitant medications |
| | AE assessment |
| | Provide available test results |

<sup>\*</sup>If indicated and/or per local standard of care

## 7.3.3 4-week Visit – Visit 6 (28 days after Visit 2)

At least four weeks after Enrollment, participants will come to the clinic for acceptability and safety evaluation for the first film, the clinician will remove any visible film, and the participant will insert a second film. Study staff will once again review instructional materials about the film and film insertion with participants prior to insertion of the second film. The second film will be the same film shape the participant was randomized to at enrollment, and film placement will be checked visually by a study clinician. If less than half of the vaginal film is proximal to introitus, participants will have the film removed and asked to try again with a new film. If less than half of the vaginal film is proximal to introitus a second time, participants will have the film removed and a third film inserted by the clinician using a speculum. Participant attempts to insert the film will be documented on the appropriate CRF. During the second month, there are no restrictions on vaginal product use or sex. Participants will be asked to provide a urine sample for a UPT, undergo HIV/STI testing and a pelvic examination, and complete an interviewer-administered acceptability questionnaire about the film.

Table 5: 4-week Visit – Visit 6 (28 days after Visit 2)

| 4-week Visit – Visit 6 (28 days after Visit 2) | |
|---|---|
| Component | Procedures |
| Administrative and Regulatory | <ul> <li>Review/update locator information</li> <li>Provide reimbursement</li> <li>Schedule next visit/contact</li> </ul> |
| Behavioral/Counseling | <ul> <li>HIV pre- and post-test counseling</li> <li>HIV/STI risk reduction counseling</li> <li>Protocol counseling (including regarding sexual partner IDI component and product use)</li> <li>Review instructional materials</li> </ul> |
| | <ul> <li>Follow-up behavioral questionnaire (acceptability and product use experiences; intravaginal practices and sexual activity)</li> <li>Post-insertion acceptability assessment</li> </ul> |
| Clinical | <ul> <li>Review/update medical and menstrual history</li> <li>Review/update concomitant medications</li> <li>Perform targeted physical examination*</li> <li>Perform pelvic examination with speculum</li> <li>AE assessment</li> <li>Treat or prescribe treatment for RTI/UTI/STIs*</li> <li>Visual examination by clinician to check vaginal film placement</li> </ul> |
| | <ul><li>Clinician film insertion assessment</li><li>Provide available test results</li></ul> |

| 4-week Visit – Visit 6 (28 days after Visit 2) | | |
|---|---|---|
| Component | | Procedures |
| | Saliva | HIV test(s) (only at sites with CLIA certification) |
| | Urine | Urine pregnancy test |
| | | Urine dipstick/culture* |
| | | HIV test(s) (not required for sites that conduct saliva testing) |
| | Blood | • CBC* |
| Laboratory | Біооц | Serum creatinine* |
| | | AST/ALT* |
| | | NAAT for GC/CT/TV |
| | | <ul> <li>Saline/KOH wet mount for candidiasis and/or BV*</li> </ul> |
| | Pelvic | Vaginal Gram stain |
| | | Vaginal swab(s) for microbiota |
| | | Vaginal pH |
| Study Product/Supplies | | Provide vaginal film for self-insertion at clinic |
| | | <ul> <li>Clinician insertion of vaginal film at clinic (only if participant fails two<br/>attempts)</li> </ul> |
| | | Offer male condoms |

<sup>\*</sup>If indicated and/or per local standard of care

## 7.3.4 Phone check-in (24-72 hours after 2nd insertion) – Visit 7

Between 24 and 72 hours after the insertion of the second film, a member of the study team will contact the study participant via telephone or SMS to assess experiences with the second vaginal film *in situ*. Participants who prefer to complete these procedures in-person may elect to do so. The staff member will ask the participant about sensation with the film in place, any experiences of leakage, and any other concerns. If conducted as a phone conversation, this is anticipated to be less than 5 minutes. If conducted as an SMS exchange, this is anticipated to be less than 5 text messages from each party. If participants raise any concerns that require more in-depth discussion, the staff member will assess the proper follow-up method.

Table 6: Phone check-in (24-72 hours after 2nd insertion) – Visit 7

| <u> </u> | |
|---|---|
| Phone check-in (24-72 hours after 2nd insertion) – Visit 7 | |
| Component | Procedures |
| Administrative and Regulatory | Provide reimbursement |
| Behavioral/Counseling | Brief behavioral assessment (concerns and comfort with film use) |

## 7.3.5 6-week Telephone Contact – Visit 8 (14 days after Visit 6)

Approximately two weeks after the second film insertion at Visit 6, the study team will contact the study participant via telephone or SMS to assess participant wellness, comfort with the film, and any concerns. Participants who prefer to complete these procedures in-person may elect to do so. Participants who report AEs or otherwise express concerns may be asked to come in for an Interim Visit, if willing, to conduct additional counseling and/or testing as needed.

Table 7: 6-week Telephone Contact – Visit 8 (14 days after Visit 6)

| 6-week Telephone Contact – Visit 8 (14 days after Visit 6) | |
|---|---|
| Component | Procedures |
| | Review/update locator information |
| Administrative and Regulatory | Provide reimbursement |
| | Schedule next visit/contact |
| Behavioral/Counseling | Brief behavioral assessment (concerns and comfort with film use) |
| Donavioral Counciling | Protocol counseling* |
| | Review/update medical and menstrual history |
| Clinical | Review/update concomitant medications |
| | AE assessment |
| | Provide available test results |

<sup>\*</sup>If indicated and/or per local standard of care

## 7.3.6 8-week Visit – Visit 9 (28 days after Visit 6)

At least four weeks after the second film insertion at Visit 6, participants will come to the clinic for acceptability and safety evaluation for the second film, and the clinician will remove any visible film. Participants will be asked to provide a urine sample for a UPT, undergo HIV/STI testing and a pelvic examination, and complete an interviewer-administered acceptability questionnaire about the film and a social harms and benefits assessment. This visit will constitute the Early Termination Visit.

Table 8: 8-week Visit – Visit 9 (28 days after Visit 6)

| 8-week Visit - | 8-week Visit – Visit 9 (28 days after Visit 6) | |
|---|---|---|
| Component | | Procedures |
| | | Review/update locator information |
| | | Provide reimbursement |
| Administrative and Regulatory | | Confirm permission to contact sexual partner for IDI (subset) and invite per site Sexual Partner Contact SOP |
| | | Schedule next visit/contact |
| | | HIV pre- and post-test counseling |
| | | HIV/STI risk reduction counseling |
| | | Protocol counseling |
| Behavioral/Counseling | | Follow-up behavioral questionnaire (acceptability and product use experiences; intravaginal practices and sexual activity) |
| | | Social harms and benefits assessment |
| | | Conduct participant IDI (subset) <sup>a</sup> |
| | | Review/update medical and menstrual history |
| | | Review/update concomitant medications |
| | | Perform targeted physical examination* |
| Clinical | | Perform pelvic examination with speculum |
| | | AE assessment |
| | | Treat or prescribe treatment for RTI/UTI/STIs* |
| | | Provide available test results |
| | Saliva | HIV test(s) (only at sites with CLIA certification) |
| Laboratory | Urine | Urine pregnancy test |
| | | Urine dipstick/culture* |

| 8-week Visit - Visit 9 (28 days after Visit 6) | |
|---|---|
| Component | Procedures |
| | HIV test(s) (not required for sites that conduct saliva testing) |
| Blood | • CBC |
| | Serum creatinine |
| | AST/ALT |
| | NAAT for GC/CT/TV |
| | <ul> <li>Saline/KOH wet mount for candidiasis and/or BV*</li> </ul> |
| Pelvic | Vaginal Gram stain |
| | Vaginal swab(s) for microbiota |
| | Vaginal pH |
| Study Product/Supplies | Offer male condoms |

<sup>\*</sup>If indicated and/or per local standard of care; a At or after Visit 9, before Visit 10

A subset of up to 35 participants will be purposively selected to complete a single explanatory IDI to provide further insight on their experiences using the placebo film and behaviors relevant to the study endpoints. The IDI Visit may occur on the same day as Visit 9 if agreed upon by the participant(s) and the study staff or may be scheduled up until Visit 10. Participants selected for the sexual partner subset IDI will be asked to confirm permission to contact their sexual partner and – if confirmed – the sexual partner will be invited per site Sexual Partner Contact SOP.

## 7.3.7 Final Telephone Contact/Study Exit Visit – Visit 10 (7 days after Visit 9)

The Final Telephone Contact will occur approximately one week after study product use has ended. The study team will contact the study participant via telephone or SMS to assess participant wellness and any concerns. Participants who prefer to complete these procedures inperson may elect to do so. This visit constitutes the Study Exit Visit (SEV) and will serve as a final safety assessment.

Table 9: Final Contact/SEV - Visit 10 (7 days after Visit 9)

| Final Contact/SEV – Visit 10 (7 days after Visit 9) | |
|---|---|
| Component | Procedures |
| Administrative and Regulatory | Review/update locator information |
| , talling all to all a regulatory | Provide reimbursement |
| | Review/update medical and menstrual history |
| Clinical | Review/update concomitant medications |
| | AE assessment |
| | Provide available test results |

#### 7.3.8 Sexual Partners – IDI Visit

Up to 30 sexual partners will be screened and enrolled to take part in a single IDI within one month of their participant partner's Visit 9. Members of the protocol team and site teams will collaboratively determine which sexual partners to contact from among those that participants have given written permission for the study team to contact. Permission to contact sexual partners will be confirmed at Visit 9, and – if confirmed – sites will contact sexual partners according to site SOP and/or local IRB/IEC guidelines. Participants may change their decision about their sexual partners' involvement at any time during the study. Selection of sexual partners to invite for an

IDI will be purposive so that characteristics/experiences of the enrolled study participant, use of film A or B, study site, and a breadth of perspectives and experiences are represented. Selection criteria and procedures will be further described in the MATRIX-002 SSP Manual. The IDI will include the following topics:

- Disclosure/knowledge/understanding of clinical study, participant's involvement in MATRIX-002, protocol restrictions on sexual activity in Month 1, and study product.
- Experiences of sex with clinical study participant during the time they were using study product.
- Perspectives and attitudes regarding monthly vaginal film use for HIV prevention.

**Table 10: IDI Visit with Sexual Partner Subset** 

| IDI Visit with Sexual Partner Subset – Screening and Enrollment Procedures | |
|---|---|
| Component | Procedures |
| | Confirm eligibility |
| | Obtain written informed consent |
| Administrative and Regulatory | Assign a unique PTID Number |
| | Collect demographic data |
| | Collect locator information |
| | Provide reimbursement for study visit |
| Behavioral | Administer brief behavioral questionnaire |
| Deliaviolai | Conduct sexual partner IDI <sup>b</sup> |

<sup>&</sup>lt;sup>b</sup> Within one month of participant Visit 9

Multiple visits may be conducted to complete all required procedures, if necessary.

## 7.4 Follow-up Procedures for Participants Who Permanently Discontinue Study Product

## 7.4.1 Participants Who Become Infected with HIV

If a participant tests positive for HIV after the Enrollment Visit, the participant will be referred to local care and treatment services and may return to the research clinic for additional counseling and other support services, as needed. Continued study participation would be of no added benefit to the participant, thus follow-up visits and procedures will be discontinued, study product use will cease, and the participant will be considered terminated from the study. An Early Termination Visit will be conducted, if the participant is willing (see Section 7.3.6). Please reference the MATRIX-002 SSP Manual for additional details.

## 7.4.2 Participants Who Become Pregnant

If a participant becomes pregnant after the Enrollment Visit, the participant will be referred to local health care services and may return to the research clinic for additional counseling, as needed. Continued study participation would be of no added benefit to the participant, thus study product use will cease, follow-up visits and procedures will be discontinued, and the participant will be considered terminated from the study. An Early Termination Visit will be conducted, if the participant is willing (see Section 7.3.6). Please reference the MATRIX-002 SSP Manual for additional details.

## 7.4.3 Participants Who Permanently Discontinue Study Product Use

Participants who permanently discontinue study product use for any clinician-initiated reason other than HIV infection or pregnancy may, after consultation with the PSRT and MATRIX-002 Management Team, have their remaining study follow-up visits and procedures discontinued. Participants will, however, be asked to complete an Early Termination Visit, if willing (see Section 7.3.6). In the event study follow-up is continued, participants will have the protocol-specified visits through SEV. Sites should contact the PSRT and management team to determine whether the participant should be followed on study and what study procedures should be completed.

Participants who permanently discontinue study product use due to an adverse event (AE) should continue to be followed in the study, if willing, until resolution (return to baseline) or stabilization of the AE is documented.

## 7.5 Interim Visits/Contacts

Interim visits/contacts (i.e., between regularly scheduled visits) may be performed as needed (e.g., participant reports an AE or social harm) at any time during the study, and any visit/contact procedures may be conducted as indicated. All interim contacts and visits will be documented in participants' study records. Refer to the MATRIX-002 SSP Manual for additional details.

## 7.6 Behavioral Evaluations

The study will address questions related to the primary, secondary, and exploratory objectives of acceptability, usability, and social harms and benefits, and both participants' and sexual partners' attitudes towards and experiences with the vaginal film. The study will assess film use facilitators and challenges experienced by participants, from the perspectives of both the participants and a subset of sexual partners. The study will also explore participants' and sexual partners' views on acceptable approaches to support study product adherence. These questions will be assessed via behavioral questionnaires and IDIs conducted by trained interviewers/facilitators. In addition, the study aims to gain further insight on:

- Product insertion
- Attitudes towards and experiences with using the vaginal film
- Perspectives on any changes in vaginal environment
- Comparisons between the two study products and comparisons to existing HIV prevention options
- Factors related to future willingness to use/recommend the vaginal film
- Sexual partner attitudes towards and experiences with the vaginal film, and their perspective of participant's attitudes and experiences

Additional questions and probes will be designed to delve further into the social and cultural norms that may play a role more broadly in product use. SMS or a phone call 24-72 hours after Visit 2 and Visit 6 will be employed as a measure to obtain information about initial experiences with vaginal film after insertion at the clinic. If a participant reports sexual activity, douching, or use of an intravaginal product, the site staff will record these behaviors on the appropriate CRF.

## **7.6.1 Quantitative Behavioral Assessments**

Participant attitudes and behaviors will be assessed throughout the study period using multiple data collection methods. Behavioral questionnaires at enrollment and during follow-up will measure key dimensions of acceptability pertinent to the vaginal film in its current phase of development alongside women's experiences in using the film during the study. In addition, behavioral questionnaires will measure vaginal practices, contraceptive use, HIV prevention behaviors, sexual behavior and relationship factors. These questionnaires will be used to assess factors correlated with placebo vaginal film acceptability and use experiences. Additionally, quantitative questionnaire data will be complemented by data captured through structured SMS and phone visits, and through IDIs with subsets of participants and sexual partners.

Table 11 outlines a summary of the assessment methods that will be used and the specific components of acceptability that will be assessed, informed by previous work and the Theoretical Framework of Acceptability as presented in Ortblad et. al.<sup>19</sup>

**Table 11: Summary of behavioral assessments** 

| Table 11: Sammary of Benavioral assessments | |
|---|---|
| Assessments and Timepoints | Acceptability components measured |
| Baseline assessment | Affective attitude, burden, opportunity costs, |
| (Visit 2) | barriers/benefits |
| Follow-up phone/SMS contacts (Visits 3-5, 7-8) | Concerns and comfort with film use |
| Follow-up assessments | Affective attitude, burden, opportunity costs, |
| (Visits 6 and 9) | overall satisfaction, usability, appropriateness, preferences, perceived barriers/benefits |
| Social harms and benefits assessment (Visit 9) | N/A |
| Participant IDI | Affective attitude, burden, satisfaction, usability, |
| (At or after Visit 9, before Visit 10) | appropriateness, perceived barriers/benefits |
| Sexual partner IDI | Affective attitude, burden, satisfaction, usability, |
| (Within one month of Visit 9) | appropriateness, perceived barriers/benefits |

## 7.6.2 Qualitative Behavioral Assessments

Two sets of IDI will be completed. The first will be conducted with a subset of participant film users who will be purposively selected and invited to complete an IDI after their second one-month period of film use. The IDI will take place at Visit 9 or scheduled after the visit and before study exit (Visit 10). Additionally, a subset of sexual partners of participants will be purposively selected to participate in an IDI, which will take place within approximately one month of Visit 9. We will explore participant experiences using the vaginal film, acceptability of shape and dependent attributes such as tactile quality of the films, and social factors influential to attitudes toward the vaginal film as a future HIV prevention option. We will also explore sexual partner views on the vaginal film and their perceptions of and experience with the film during sexual activity. IDIs will be conducted separately with participants and their sexual partners to assess these topics. IDIs will include, but not be limited to, the following topics:

- Descriptions of film insertion practices
- Main challenge(s) encountered with film use, especially during sex
- Potential changes to the film
- Other factors (e.g., situational, relationship, trial-specific, social/cultural/economic, sex and menstruation related, vaginal practices) influencing film acceptability and use experience
- Sexual partner attitudes towards and experiences with the vaginal film, and their perspective of participant's attitudes and experiences

Semi-structured IDI guides will be developed by qualified social scientists and administered by qualified interviewers. Guides will contain key research questions relating to the main topics of interest and suggested probes. Interviews and discussion sessions will be audio-recorded and transcribed.

## 7.7 Protocol Adherence Counseling

Participants will receive protocol counseling upon enrollment into the study (Visit 2) and at Visit 6 as appropriate to the visit. Study staff will document administration of study product and that the counseling was provided. Contraception counseling will be provided to participants of childbearing potential at all clinic visits beginning at Screening. Protocol adherence counseling will be provided at all clinic visits beginning at Screening, except SEV. Counseling will be provided by different site staff than those conducting the behavioral assessments when feasible, in accordance with standard study methods and as specified in site SOPs. Counseling also will include reminders regarding concomitant medication, sexual activity, intravaginal product use and practices, and behavioral restrictions during study participation as specified in Section 6.7.

## 7.8 Clinical Evaluations and Procedures

## Physical Examination and Medical History

The full physical examination will include the following assessments:

- Vital signs
  - Blood pressure
- Measurements of weight and height
- General appearance
- Cardiac exam
- Respiratory exam
- Abdomen

Participants will be asked about medications/therapies at every visit, including Screening. Study staff will ask about adverse events at all visits beginning at Enrollment. A full physical examination will be completed by a clinician at Screening. Thereafter, a targeted physical examination will be performed to assess any complaints or symptoms with which the participant presents at the follow-up visits as clinically indicated.

#### Pelvic Examination

Pelvic exams will be performed using visual inspection of external genitalia and using a speculum for examination of the cervix and vagina, assessment of film persistence, and insertion of film (if

participant fails first two attempts). Bimanual exam may be performed as needed (required at Screening Visit). Pelvic exams will be conducted at Screening, Enrollment, and Visits 6 and 9 for vaginal microenvironment specimen collection and as indicated based on participant reports. Cervicovaginal fluid (CVF) will be collected using swabs.

Additional clinical assessments/procedures may be performed at the discretion of the examining clinician in response to symptoms or illnesses present at the time of the exam/procedure.

## 7.9 Laboratory Evaluations

#### Local Laboratory

- Saliva (only at sites with CLIA certification)
  - HIV test(s)
- Urine
  - Urine pregnancy test
  - Urine dipstick/culture (as indicated, per local standard of care)
- Blood
  - HIV test(s) (not required for sites that conduct saliva testing)
  - o CBC
  - Serum creatinine
  - AST/ALT
  - Syphilis serology
- Pelvic
  - NAAT for GC/CT/TV
  - Pap test (if indicated [if participant is unable to provide documentation of a normal Pap test within 3 years prior to enrollment])
  - KOH wet mount for candidiasis and/or BV (if indicated)
  - Vaginal pH

## Designated Laboratory

- Blood
  - Plasma for archive
- CVF
  - Gram Stain for Nugent Scoring
  - Microbiota

Only Local Laboratory test results will be provided to the participant. Once all required study analyses of collected specimens are complete, any remaining samples may be shipped to Pitt/MWRIF for use in study-related quality assurance and quality control testing. If study samples will be used for assay validation or proficiency testing that is not study related, all participant identifiers (PTID) will be removed from the samples prior to use. Specimens obtained from participants who do not consent to long term storage will not be used for assay validation or proficiency testing purposes and will be destroyed when all protocol-specified testing has been completed.

## 7.10 Specimen Management

Study sites will adhere to the standards of good clinical laboratory practice, in accordance with the MATRIX-002 SSP Manual and site SOP for proper collection, processing, labeling, transport, and storage of specimens. Specimen collection, testing, and storage at the site laboratories will be documented when applicable using the Laboratory Data Management System (LDMS). In cases where laboratory results are not available due to administrative or laboratory error, or out of range and the site IoR/designee determines reasonable to repeat, the site is permitted to re-draw specimens. No genetic testing (limited or genome-wide) is planned on leftover samples that are stored for the purposes of future research.

## 7.11 Laboratory Oversight

All laboratories participating in this study will adhere to MATRIX's Laboratory Policy (www.matrix4prevention.org).

#### 7.12 Biohazard Containment

As the acquisition of HIV and other blood-borne pathogens can occur through contact with contaminated needles, blood, and blood products, appropriate blood and secretion precautions will be employed by all personnel in the drawing of blood and shipping and handling of all specimens for this study as recommended by the US Centers for Disease Control and Prevention (CDC), National Institutes of Health (NIH), and other applicable national regulatory authorities. All biological specimens will be transported using packaging mandated by Code of Federal Regulations (CFR) 42 Part 72. All dangerous goods materials, including diagnostic specimens and infectious substances, must be transported according to instructions detailed in the International Air Transport Association (IATA) Dangerous Goods Regulations. Biohazardous waste will be contained according to institutional, transportation/carrier, and all other applicable regulations.

## 8 ASSESSMENT OF SAFETY

## 8.1 Safety Monitoring

Site IoRs/designees are responsible for continuous close safety monitoring of all study participants, and for alerting the Protocol Team if unexpected concerns arise. A sub-group of the Protocol Team, including the Protocol Co-Chairs, Protocol Safety Physician, Clinical Research Manager(s) (CRM), and Pitt/MWRIF representatives will serve as the PSRT. The Clinical Data Manager(s) (CDM) prepares routine AE and clinical data reports for review by the PSRT, which meets via conference call approximately once per month or more frequently as needed throughout the period of study implementation to review safety data, discuss product use management, and address any potential safety concerns.

## 8.2 Clinical Data and Safety Review

A multi-tiered safety review process will be followed for the duration of this study. The site IoRs/designees are responsible for the initial evaluation and reporting of safety information at the participant level and for alerting the PSRT if unexpected concerns arise. Participant safety is also monitored through a series of routine reviews conducted by the PSRT and (if applicable) study sponsors. Additional reviews may be conducted at each of these levels as dictated by the occurrence of certain events.

The CDM(s) will review incoming safety data on an ongoing basis. Events identified as questionable, inconsistent, or unexplained will be queried for verification. To ensure prompt review of AEs of concern (e.g., serious adverse events [SAE] and Related Grade 3+ AEs), such AE reports submitted in the clinical database will be forwarded to the PSRT for review within 72 hours of entry.

The PSRT will meet approximately every month, or as needed, via conference call to review clinical data reports generated by the CDM(s). The content, format and frequency of the clinical data reports will be agreed upon by the PSRT and the CDM(s) in advance of study implementation. In addition to the routine safety data reviews, the PSRT will convene on an ad hoc basis to make decisions regarding the handling of any significant safety concerns. If necessary, experts external to MATRIX representing expertise in the fields of microbicides, biostatistics, HIV acquisition and medical ethics may be invited to join the PSRT safety review. A recommendation to pause or stop the trial may be made by the PSRT at this time or at any such time that the team agrees that an unacceptable type and/or frequency of AEs has been observed.

The Independent Safety Physician (ISP) will review participant safety data as part of their regular reviews (see Section 10.6.1), since no Data and Safety Monitoring Board (DSMB) oversight is planned for MATRIX-002. These reviews will take place approximately every 3 months, or as needed. The ISP will be an independent investigator(s) with no interest (financial or otherwise) in the outcomes of this study. At the time of these reviews, or at any other time, the ISP or PSRT may convene a panel (composed of the ISP, PSRT and protocol statistician[s]) to review study findings. This panel may recommend that the study proceed as designed, proceed with design modifications, or be discontinued. If at any time a decision is made to discontinue enrollment and/or study product use in all participants, Pitt/MWRIF will notify USAID and (as necessary) relevant regulatory autorities, and Site IoRs/designees will notify the responsible IRBs/IECs expeditiously per local guidelines.

## 8.3 Adverse Events Definitions and Reporting Requirements

#### 8.3.1 Adverse Events

An AE is defined as any untoward medical occurrence in a clinical research participant administered an investigational product and which does not necessarily have a causal relationship with the investigational product. As such, an AE can be an unfavorable or unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of an investigational product, whether or not considered related to the product. This definition is applied to all study participants and is applied beginning at the time of

enrollment (i.e., once a participant is randomized). The term "investigational products" for this study refers to the two placebo vaginal films A and B.

Study participants will be provided instructions for contacting the study site to report any untoward medical occurrences they may experience. In cases of potentially life-threatening events, participants will be instructed to seek immediate emergency care. Where feasible and medically appropriate, participants will be encouraged to seek evaluation where a study clinician is based, and to request that the clinician be contacted upon their arrival. With appropriate permission of the participant, whenever possible, records from all non-study medical providers related to untoward medical occurrences may be obtained and required data elements will be recorded on study CRF. All participants reporting an untoward medical occurrence should be followed clinically until the occurrence resolves (returns to baseline) or stabilizes.

Study site staff will document in source documents and in the study database all AEs reported by or observed in enrolled study participants regardless of severity and presumed relationship to study product. AE severity will be graded per the DAIDS Table for Grading Adult and Pediatric Adverse Events, Corrected Version 2.1, July 2017 and/or Addenda 1 (Female Genital Grading Table for Use in Microbicide Studies [Dated November 2007]).

Asymptomatic BV and asymptomatic candidiasis will not be reportable AEs but will be captured on the appropriate study CRF. Bleeding at the time of speculum insertion/removal and/or cervicovaginal specimen collection that is judged by the clinician to be within the range of normally anticipated for that procedure, will not be reportable as an AE. Bleeding that is judged by the clinician to be due to contraception use will also not be reportable as an AE.

For any SAEs that are continuing at a participant's study exit visit, the IoR/designee must establish a clinically appropriate follow-up plan for the AE. At a minimum, the SAE must be re-assessed by study staff 30 days after the participant's study exit visit; additional evaluations also may take place at the discretion of the IoR/designee.

The same approach must be taken for any AEs that are found to have increased in severity to Grade 3 or higher at the study exit visit. For those AEs requiring re-assessment, if the AE has not resolved or stabilized at the time of re-assessment, study staff should continue to re-assess the participant at least once per month while the study is ongoing. After the study has ended, all AEs requiring re-assessment should be re-assessed at least once within the 30 days after the study end date.

Grade 1 and Grade 2 AEs classified as "related" to study product or procedures still ongoing at study exit require follow up by the study team at least once within 30 days of study exit.

The PSRT may advise study staff as to whether any additional follow-up may be indicated on a case-by-case basis. For AEs that are re-assessed after study exit, information on the status of the AE at the time of re-assessment will be recorded in source documents only — no updates should be made to AE CRFs based on the re-assessments.

#### 8.3.2 Serious Adverse Events

As per the International Council for Harmonization of Technical Requirements for Pharmaceuticals for Human Use Good Clinical Practice Guidance (ICH E6; https://www.ich.org/page/efficacyguidelines), SAEs are defined as AEs occurring at any dose that:

- Results in death
- Is life-threatening
- Results in persistent or significant disability/incapacity
- Is a congenital anomaly/birth defect
- Requires inpatient hospitalization or prolongation of existing hospitalization

NOTE: Per ICH SAE definition, hospitalization itself is not an AE, but is an outcome of the event. Thus, hospitalization in the absence of an AE is not regarded as an AE. The following are examples of hospitalization that are not considered to be AEs:

- o Protocol-specified admission (e.g., for procedure required by study protocol)
- Admission for treatment of target disease of the study, or for pre-existing condition (unless it is worsening or increases in frequency of hospital admissions as judged by the clinical investigator)
- Diagnostic admission (e.g., for a work-up of an existing condition such as persistent pretreatment lab abnormality)
- Administrative admission (e.g., for annual physical)
- Social admission (e.g., placement for lack of place to sleep)
- Elective admission (e.g., for elective surgery)

Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.

## **8.3.3 Adverse Event Relationship to Study Product**

Relatedness is an assessment made by a study clinician of whether or not the event is related to the study agent. The relationship categories that will be used for this study are:

- Related: There is a reasonable possibility that the AE may be related to the study agent(s)
- Not Related: There is not a reasonable possibility that the AE is related to the study agent(s)

## 8.4 Pregnancy and Infant Outcomes

Pregnant women are excluded from this study. A participant who becomes pregnant during the study will have study product discontinued and will be terminated from the study. Please see Section 9.7 for additional details.

## 8.5 Regulatory Requirements

AEs reported on CRFs will be included in reports to the applicable national drug regulatory authorities (DRA) in accordance with DRA requirements. Site IoRs/designees also will submit AE information and any other relevant safety information to their IRB/IEC in accordance with IRB/IEC requirements.

## 8.6 Social Harms Reporting

Although study sites will make every effort to protect participant privacy and confidentiality, it is possible that participants' involvement in the study could become known to others and that social harms may result. For example, participants could be treated unfairly, or could have problems being accepted by their families, partners and/or communities. Social harms that are judged by the IoR/designee to be serious or unexpected will be reported to the PSRT and responsible site IRB/IEC according to their individual requirements. In the event that a participant reports social harm, every effort will be made by study staff to provide appropriate care and counseling to the participant, and/or referral to appropriate resources for the safety of the participant as needed. While maintaining participant confidentiality, study sites may engage their community advisory boards (CABs) in exploring the social context surrounding instances of social harm. To mitigate one possible source of social harms, each site will carefully explain to eligible participants the potential consequences of enrolling their sexual partner (e.g., disclosure of study involvement and/or film use) prior to contacting the partner.

## 9 CLINICAL MANAGEMENT

Guidelines for clinical management and permanent discontinuation of study product are outlined in this section. Permanent discontinuation of study product will be defined as not having the second film inserted at Visit 6. In general, the IoR/designee has the discretion to hold study product at any time if s/he feels that continued product use would be harmful to the participant or interfere with treatment deemed clinically necessary. Unless otherwise specified below, the IoR/designee should immediately consult the PSRT for further guidance on resuming study product during second month of product use (if product discontinuation occurs during first month of product use) or progressing to permanent discontinuation of study product and early study termination. The IoR/designee will document all permanent discontinuations on applicable CRFs.

## 9.1 Grading System

AE severity grading is described in Section 8.3.1.

#### 9.2 Dose Modification Instructions

No dose modifications will be undertaken in this study.

## 9.3 General Criteria for Permanent Discontinuation of Study Product

A participant will be <u>permanently discontinued</u> from product use by the IoR/designee for any of the following reasons:

- A reactive rapid HIV test.
- Pregnancy or breastfeeding.
- Allergic reaction to the study product(s)/drug(s).
- Reported use of or need for PrEP or PEP. Participants who experience a known or potential
  HIV exposure during study participation or have a recognized risk of exposure and thus
  need PEP or PrEP will have study product permanently discontinued and will be referred
  for PEP or PrEP initiation. Those who need PEP will be encouraged to start it as quickly as
  possible and within 72 hours of potential exposure. Since continued study follow-up would
  be of no benefit following permanent discontinuation of study product use, these
  participants will be exited from the study.
- Non-therapeutic injection drug use.
- Participant develops a Grade 3 Related or Grade 4 AE.
- Participant is unable or unwilling to comply with required study procedures, or otherwise might be put at undue risk to their safety and well-being by continuing product use, according to the judgment of the IoR/designee.

The IoR/designee must consult the PSRT on all discontinuations instituted at their discretion for further guidance on resuming product use during second month of product use (if product discontinuation occurs during first month of product use) or progressing to permanent discontinuation of study product and early study termination.

## 9.4 Permanent Discontinuation in Response to Observed Adverse Events

## **Grade 1, Grade 2 and Grade 3 Unrelated**

Unless specifically addressed in Section 9.5 below, a participant who develops a Grade 1 or 2 AE, regardless of relationship to study product, may continue product use. Participants who develop a Grade 3 AE that is judged by the IoR/designee to be unrelated to study product may also continue product use. If the IoR/designee opts to discontinue study product, the PSRT must be notified.

#### **Grade 3 Related and Grade 4**

Study product must be permanently discontinued and the PSRT notified for participants who develop a Grade 3 Related AE or a Grade 4 AE.

## 9.5 Other Clinical Findings

A thorough evaluation of genital complaints is expected in the context of this study; however, syndromic management of genital symptoms is acceptable while awaiting laboratory results if such practice is in line with the local standards of care. Observed single dose treatment should be provided whenever possible, per clinician discretion. When clinically appropriate, investigators should use oral or parenteral medications when at all possible.

Product use need not be held in the event of an STI/RTI requiring treatment, unless other permanent discontinuation guidelines apply. Should the IoR/designee determine that a

permanent discontinuation is warranted due to an STI or RTI, consultation with the PSRT is required. The IoR/designee should manage STI/RTI per local guidelines or current WHO guidelines, available at http://www.who.int/en/. Test for cure is not required after treatment of asymptomatic STIs.

If a suspected finding is reported by the participant between scheduled visits, an interim visit may be scheduled at the discretion of the site investigator.

#### 9.6 HIV Infection

HIV testing will be performed at designated study visits. Potential participants who test positive for HIV during Screening or Enrollment will not be enrolled in the study but will be referred to HIV care and management. Enrolled participants who test positive for HIV will have study product and all follow-up visits discontinued, and will be considered terminated from the study as per Section 7.4.1. Participants identified as infected with HIV are managed or referred for management according to the local standard of care. Guidance regarding management and referral for participants confirmed to be HIV-positive can be found in Section 13.10. Sites will not be responsible for paying for HIV-related care.

## 9.7 Pregnancy

Pregnancy testing will be performed at designated study visits and participants will be encouraged to report all signs or symptoms of pregnancy to study staff. The IoR/designee will counsel any participant who becomes pregnant according to site SOPs. The IoR/designee also will refer the participant to all applicable services; however, sites will not be responsible for paying for pregnancy-related care. A participant who becomes pregnant during the course of the study will have study product and all follow-up visits discontinued, and will be considered terminated from the study as per Section 7.4.2.

## 9.8 Criteria for Early Termination of Study Participation

Participants may voluntarily withdraw from the study for any reason at any time. IoRs/designees also may withdraw participants from the study to protect their safety and/or if they are unwilling or unable to comply with required study procedures. Sites must notify the PSRT immediately of any such instances. Participants also may be withdrawn if Pitt/MWRIF, USAID, MATRIX, government or regulatory authorities, including the Office for Human Research Protections (OHRP), or site IRB/IEC/DRA terminate the study prior to its planned end date. Every reasonable effort is made to complete a final evaluation of participants who withdraw or are withdrawn from the study prior to completing follow-up (see details regarding the Early Termination Visit in Section 7.3.6). Study staff members will record the reason(s) for all withdrawals in participants' study records.

## 10 STATISTICAL CONSIDERATIONS

## 10.1 Overview and Summary of Design

MATRIX-002 is a two-arm, randomized, multi-center trial to assess acceptability, safety and usability of two placebo prototype films when administered vaginally once monthly for two months. The primary objective of MATRIX-002 is to assess the acceptability of two placebo film types (A and B) administered vaginally once monthly for two months, with the overall goal of drawing on findings across primary, secondary and exploratory endpoints to inform design of drug-loaded vaginal film.

## **10.2 Study Endpoints**

## **Primary endpoints**

## Acceptability

• Participant ratings of overall satisfaction with using the placebo vaginal films.

## **Secondary endpoints**

## Safety

• Proportion of participants with genitourinary Grade 2 or higher Adverse Events deemed related to study product.

## **Usability**

• Proportion of participants with clinically assessed proper insertion (more than half of the vaginal film proximal to introitus).

## **Exploratory endpoints**

## Participant acceptability, attitudes and experiences

- Participant responses to quantitative acceptability assessments and IDI questions. Multiple dimensions will be explored, including:
  - Vaginal film attributes, including acceptability (e.g., ease of insertion, burden, perceived effectiveness of film as delivery form) and preferences
  - Experience and comfort with inserted vaginal film (e.g., expulsions, leakage, awareness of film during daily activities)
  - Experience during sex and menses
  - Vaginal practices and concomitant vaginal product use while using vaginal film
  - o Perception of sexual partners' attitudes towards vaginal film
  - Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option
  - o Interest in using vaginal film as a future HIV prevention option

## **Sexual partner attitudes and experiences**

- Sexual partner responses during IDI related to:
  - Vaginal film attributes, including acceptability and preferences
  - o Perception of participant's experience using the vaginal film during the study

- Physical sensation of the participant's vaginal film use during sex (as relevant)
- Perceived benefits and concerns/challenges with the vaginal film as a future HIV prevention option

## **Vaginal microenvironment**

- Change from baseline in vaginal pH following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in quantity of selected vaginal microbiota following film use during the two study phases (i.e., with and without sexual abstinence requirement).
- Change from baseline in Nugent score following film use during the two study phases (i.e., with and without sexual abstinence requirement).

## Social harms and social benefits

- Participant self-report of social harms (i.e., non-clinical adverse consequences of study participation or product use that may manifest in social, psychological or physical ways).
- Participant and sexual partner self-report of social benefits (e.g., positive consequences of product use disclosure such as self-confidence, improved communication with intimate partner) resulting from vaginal film use and/or study participation.

## **10.3 Sample Size and Power Calculations**

MATRIX-002 will enroll approximately 100 evaluable participants (i.e., participants who complete Visit 6), with approximately 20 participants per site. Participants will be randomized to the 2 study arms in a 1:1 ratio, allocating 50 women per arm. In light of the short study duration and the teams' previous experiences conducting similar research with the study's target population, we anticipate 5% LTFU. Therefore, we expect approximately 95 participants (45-48 per arm) will complete the study. A subset of up to 35 study participants will complete an IDI after the 2<sup>nd</sup> period of film use. We will enroll up to 30 sexual partners to complete an IDI after the participant completes the 2<sup>nd</sup> period of film use.

Note: Replacement participants will be considered in consultation with study leadership if LTFU is higher than expected.

Table 12 presents the range of potential detectable effect sizes reflecting differences in primary, secondary and exploratory endpoints of the two study products assuming 80% power, two-sided  $\alpha$ =0.05, varying standard deviations or marginal probabilities, a sample size of 100, and 5% LTFU.

The primary acceptability endpoint will be measured at Visits 6 and 9. Secondary endpoints will be assessed cumulatively to calculate an overall proportion experiencing the outcome (e.g., AE). The usability of the vaginal film will be determined by clinician-observed and participant-reported measures (e.g., ease of insertion, number of attempts). Exploratory acceptability endpoints will be collected at Visits 6 and 9. In addition, interim data on experience using the placebo vaginal film will be collected 24-72 hours after each film insertion and again 1 week (1st use period only) and 2 weeks after each film insertion via SMS or telephone.

Table 12: Range of potential effect sizes for each endpoint

| Continuous outcomes: effect size is difference in means | | | |
|---|---|---|---|
| Endpoint | Endpoint type | Standard deviation | Minimum detectable |
| | | | difference |
| Overall satisfaction | Primary: Acceptability | 0.5 – 3.0 | 0.29 – 1.75 |
| (Likert scale 1-10) | | | |
| Likelihood of future use | Exploratory: Acceptability | 0.4 - 1.0 | 0.23 - 0.59 |
| (Likert scale 1-4) | | | |
| Binary outcomes: effect size is risk difference | | | |
| Endpoint | Endpoint type | Marginal probabilities | Minimum detectable |
| Litapolite | спаропіс суре | Platginal probabilities | difference |
| Adverse events | Safety | 0.10 - 0.30 | 0.24 - 0.29 |

## **Qualitative data collection**

Participant experiences: Up to 35 study participants will be purposively selected and invited to complete an IDI at Visit 9 or before study exit.

Sexual partner attitudes and experiences: Up to 30 sexual partners will be invited to provide insights into their attitudes and experiences through IDIs.

An overall sample of 30 IDIs per group is estimated to provide sufficient opportunity to reach saturation in the qualitative data on key topics. An estimated 6 IDIs per site per group is expected to provide sufficient opportunity for any variation on key topics based on geographic location. Participants will be purposively selected for invitation to an IDI based on vaginal film assignment (A or B) and other characteristics or experiences while using the study product. Sexual partners will be purposively selected for invitation to the IDI based on permission provided by the clinical study participant, key experiences reported by the clinical study participant, and partner interest/availability.

#### **10.4 Randomization Procedures**

Participants will be randomized in a 1:1 ratio to the two study arms (Film A or Film B), stratified by study site. The randomization scheme and procedures will be generated and maintained by the MWRI statistical team that will conduct and coordinate the randomization procedures.

## 10.5 Participant Accrual, Follow-up and Retention

We anticipate participant accrual to take place over a period of approximately 3-6 months. Each participant enrolled will be followed for a period of approximately 2 months.

## 10.6 Data and Safety Monitoring and Analysis

## 10.6.1 Study Monitoring

No DSMB oversight is planned for this study. The MATRIX Clinical Trials Hub will conduct interim reviews of study progress, including rates of participant accrual, retention, completion of primary and secondary endpoint assessments, and study or laboratory issues. The ISP will conduct interim review of incident AEs. These reviews will take place approximately every three months, or as needed. At the time of these reviews, or at any other time, the ISP or PSRT may convene a panel

(composed of the ISP, PSRT and protocol statistician[s]) to review study findings. This panel may recommend that the study proceed as designed, proceed with design modifications, or be discontinued. Safety monitoring will be done by the PSRT.

## 10.6.2 Primary Analysis(es)

All participants randomized into the study who complete Visit 6 will be included in the primary analysis.

When the use of descriptive statistics to assess group characteristics or differences is required, the following methods will be used: for categorical variables, the number and percent in each category; for continuous variables, the mean, median, standard deviation, quartiles and range (minimum, maximum). Overall and within-treatment group assessment of the change from the baseline measurement to a follow-up measurement will be analyzed using McNemar's test (for categorical response variables) or the paired t-test or Wilcoxon signed-ranks test (for continuous variables). When using formal testing to assess endpoint differences between users of Film A or Film B, the following methods will be used: for binomial response variables, chi-square tests and logistic regression (or exact testing methods); for continuous variables, t-tests and linear regression or nonparametric methods if data are non-Normal.

To assess the adequacy of the randomization, participants in each arm will be compared for baseline characteristics including demographics and laboratory measurements using descriptive statistics. Due to the small sample size, formal comparisons will not be done.

We will calculate overall estimates for mean satisfaction rating at Visit 9 (Likert 10-point scale) and by study arm to permit comparisons between Film A and Film B. We will test for difference in mean overall satisfaction rating at Visits 6 and 9 (Likert 10-point scale) between Film A and Film B using a two-sided t-test (primary endpoint). A nonparametric test will be used if normality assumptions are not met. Analyses will examine sociodemographic and behavioral correlates of acceptability rating (i.e., satisfaction) using linear regression models with robust standard errors.

## 10.6.3 Secondary and Exploratory Analyses

## Safety

All visits in which participants have been exposed to the study products will be included in the analysis of safety. Secondary intent to treat analyses may also be performed. To assess genitourinary safety, the number and percentages of participants experiencing each safety endpoint (see Section 10.2) will be tabulated by study arm as well as the total number of safety endpoints experienced in each arm. Each participant will contribute once in each category (i.e., only for the highest severity AE for each participant) for the calculation of event rates. Exact binomial confidence intervals will be calculated for each safety endpoint for each arm.

#### Usability

Usability, participants' ability to insert the film correctly, will be examined by calculating the proportion of participants who correctly inserted the film on the first attempt (and after two attempts). This will be examined by study arm and overall. Changes in ability to insert the film correctly will examine this measure at V6 and V9, by study arm and overall.

## **Exploratory Acceptability Assessment**

In addressing the exploratory acceptability objective, we will compare ratings of acceptability measures reflecting distinct components of the acceptability framework and related dimensions by study arm. Acceptability endpoints will be summarized by assessment time point (Visits 2, 6, and 9) using descriptive statistics (e.g., frequencies, means), as appropriate. For example, we will examine the level of interest in future use of the film as an HIV prevention option overall and by study arm. We will also examine responses over time (e.g., ratings of anticipated comfort prior to initial film insertion, after first month of film use, and after second month of film use), assessing whether they changed with increased experience with product insertion. In addition, analyses will examine sociodemographic and behavioral correlates of acceptability endpoints using linear regression models with robust standard errors (for rating outcomes) and using multivariable logistic regression for dichotomous outcomes such as willingness to use (e.g., disinterest in future use).

## Participant and Sexual Partner Attitudes and Experiences

Qualitative data will be audio-recorded, processed, and coded for qualitative analyses, using Dedoose or a similar qualitative software. Data coding will be used as a primary analytical approach for data reduction, that is, to summarize, extract meaning, and condense the data. Transcripts will be coded first through descriptive coding for key themes and topics, using a preliminary codebook. Additional codes will be identified through an iterative process of reading the textual data to identify emergent themes, and the codebook will be modified accordingly. In addition to descriptive codes, inductive codes, which achieve a greater level of abstraction, will be used to start linking themes and topics together in order to explore the relationship between socio-contextual factors and product use experiences. Whenever possible, we will also compare study sites and explore differences or similarities due to different socioeconomic, cultural and geographical contexts. The analysis will be done by the investigative team, working interactively through emails, and regular phone or face-to-face meetings. The findings and interpretations of the data will be critically discussed until there is group consensus on the dominant themes and meanings contained in the data.

## 10.6.4 Missing Data

In any situation with missing data, appropriate secondary analyses will be performed to adjust for variables that may be related to the missingness mechanism. If missing data rates are higher than 10%, covariates that are related to missingness in likelihood-based regression models will be included. Sensitivity analyses to assess the potential impact of the missing data will also be performed. These analyses will include imputing the data under the most extreme scenarios of information missingness, such as assuming everyone missing has an extreme value of the missing variable, and less informative imputation approaches.

## 11 DATA HANDLING AND RECORDKEEPING

## 11.1 Data Management Responsibilities

Data collection tools will be developed by the CDM(s) in conjunction with the protocol team. Quality control and data integrity are managed manually and systematically with reports and

queries routinely generated and provided by the CDM(s) to the study sites for verification and resolution. As part of the study activation process, each study site will identify all CRFs to be used as source documents. Study CRF data will be entered and managed using REDCap, a data management system compliant with the International Council on Harmonization (ICH) Good Clinical Practices (GCP) and US CFR guidelines for electronic data capture.

Transcriptions of interviews will be generated in the field and electronically transferred to RTI International using a secure File Transfer Protocol site, where they will be uploaded and managed using a qualitative software package. RTI International will act as a hub and manage all qualitative data for the study. A convention for file naming will be developed, and all data will be labeled according to this process. RTI International will save all versions of all files on a secure, password-protected server in the US.

## 11.2 Source Documents and Access to Source Data/Documents

All study sites will maintain source data/documents in accordance with MATRIX's Good Documentation Practice (GDP) guidelines (www.matrix4prevention.org).

Each IoR/designee will maintain, and store securely, complete, accurate and current study records throughout the study. In accordance with U.S. regulations, IoRs/designees will maintain all study documentation for at least three years after completion of the study.

Study records must be maintained on site for the entire period of study implementation. Thereafter, instructions for record storage will be provided by Pitt/MWRIF. No study records may be moved to an off-site location or destroyed prior to receiving approval from Pitt/MWRIF.

## 11.3 Quality Control and Quality Assurance

Study sites will conduct quality control and quality assurance procedures in accordance with MATRIX's Quality Management Plan (www.matrix4prevention.org).

## 12 CLINICAL SITE MONITORING

Study monitoring will be carried out by the African Clinical Research Organisation (ACRO) for the African sites and by the University of Pittsburgh Education and Compliance Support for Human Subject Research (ECS-HSR) for the US site. Study monitors will do the following:

- Review informed consent forms, procedures, and documentation.
- Assess compliance with the study protocol, Good Clinical Practices (GCP) guidelines, and applicable regulatory requirements (US and non-US), including US Code of Federal Regulations (CFR) Title 45 Part 46 and Title 2 Parts 200 and 225.
- Perform source document verification to ensure the accuracy and completeness of study data.
- Verify proper collection and storage of biological specimens.
- Verify proper storage, dispensing, and accountability of investigational study products.

• Assess implementation and documentation of internal site quality management procedures.

Monitoring visits may be conducted on-site or remotely. Remote visits may include remote source document verification using methods specified for this purpose. Remote monitoring visits may be performed in place of or in addition to onsite visits to ensure the safety of study participants and data integrity.

For on-site visits, the IoR/designee will allow study monitors to inspect study facilities and documentation (e.g., informed consent forms, clinic and laboratory records, other source documents, CRFs), as well as observe the performance of study procedures. The IoR/designee also will allow inspection of all study-related documentation by authorized representatives of MATRIX, Pitt/MWRIF, USAID, OHRP, IRB/IEC and other local, US, or international regulatory authorities. A site visit log will be maintained at the study site to document all visits.

## 13 HUMAN SUBJECTS PROTECTIONS

Site investigators will make efforts to minimize risks to participants. Participants and study staff members will take part in a thorough informed consent process. Before beginning the study, IoRs/designees will have obtained IRB/IEC approval. IoRs/designees will permit audits by USAID, OHRP, MATRIX, IRB/IEC, and other local, US, or international regulatory authorities or any of their appointed agents.

Changes to this protocol may be implemented by investigators prior to IRB/IEC approval, if those changes are required to eliminate apparent immediate hazards to the study participant; see 45 CFR 46.108(a)(3)(iii) under the 2018 Requirements (https://www.ecfr.gov). These changes must be documented as Protocol Deviations and reported to the Protocol Team and IRB/IEC as soon as possible; see ICH E6(R2), Good Clinical Practice, Section 4.5.4 (https://www.fda.gov/science-research/clinical-trials-and-human-subject-protection/ich-guidance-documents). In the event of a public health emergency, investigators should adhere to the recommendations of their local institutions, IRB/IEC and local health departments. When conflicts exist between local directives, MATRIX, Protocol Team and/or USAID policies or guidance, sites should follow the requirement that is most protective of study participants and site staff.

## 13.1 Institutional Review Boards/Ethics Committees

Each participating institution will be responsible for assuring that this protocol, the associated site-specific informed consent forms (ICF), and study-related documents (such as participant education and recruitment materials) are reviewed by the IRB/IEC responsible for oversight of research conducted at their study site and by applicable national DRA. Any amendments to the protocol must be approved by the responsible IRBs/IECs and (if applicable) national DRA prior to implementation.

Subsequent to the initial review and approval, the responsible IRBs/IECs must review the study at least annually. Each IoR/designee will make safety and progress reports to their IRB/IEC and (if applicable) to their national DRA at least annually and within three months after study

termination or completion. These reports will include the total number of participants enrolled in the study, the number of participants who completed the study, all changes in the research activity, and all unanticipated problems involving risks to human subjects or others. In addition, the results of all safety reviews of the study will be provided to the IRBs/IECs and (if applicable) national DRA.

## 13.2 Protocol Implementation

Prior to implementation of this protocol, and any subsequent full version amendments, each site must have the protocol and the protocol consent forms approved, as appropriate, by their local IRB/IEC and any other applicable regulatory entities. Upon receiving final approval, sites will submit copies of all relevant protocol/amendment documents (i.e., IRB/IEC approval letters with a detailed list of approved documents, approved ICF documents, etc.) to the MATRIX Clinical Trials Hub Regulatory team.

The MATRIX CRM(s) will review the submitted document packet to ensure receipt of all required protocol/amendment documents prior to study activation at the sites. Sites will receive a Study Activation Notification from the MATRIX CRM(s) that indicates successful completion of the protocol readiness process. A copy of the Study Activation Notification should be retained in the site's regulatory files.

Upon receiving final IRB/IEC and any other applicable approval(s) for an amendment, activated sites should implement the amendment immediately but are still required to submit copies of all relevant amendment documents to the MATRIX Clinical Trials Hub Regulatory team.

## **13.3 Study Coordination**

Study implementation will be directed by this protocol, which may not be amended without prior written approval from the Protocol Co-Chairs and Protocol Team representatives from MATRIX, Pitt/MWIF and USAID. Study implementation will also be guided by a common SSP Manual that provides further instructions and operational guidance on conducting study visits; data and forms processing; specimen collection, processing, and shipping; AE assessment, management and reporting; dispensing study products and documenting product accountability; and other study operations. Standardized study-specific training will be provided to sites by the MATRIX CRM(s) and other designated members of the Protocol Team.

Close coordination between protocol team members is necessary to track study progress, respond to queries about proper study implementation, and address other issues in a timely manner. The PSRT will address issues related to study eligibility and AE management and reporting as needed to assure consistent case management, documentation, and information-sharing across sites. Rates of accrual, adherence, follow-up, and AE incidence will be monitored closely by the team as well as the ISP and the MATRIX Clinical Trials Hub.

#### 13.4 Risk Benefit Statement

## 13.4.1 Risks

## General

HIV and STI testing may make the participant feel anxious regardless of the test results. Counseling and testing for HIV and other STIs may cause worry and discomfort by learning more about risk for those conditions. A participant may become worried, sad or depressed after finding out that they have HIV or an STI. Trained study staff will be available to help participants deal with these feelings.

Finding out their HIV status could also cause problems between participants and their partners, family, or friends. Participants also could have problems in their partner relationships associated with study-required abstinence. The study staff will provide counselling and referral for support and/or care where required.

Participation in clinical research includes the risk of loss of confidentiality and discomfort with the personal nature of questions when discussing sexual behaviors. Study staff will make every effort to protect participant privacy and confidentiality during the study visits. Visits will take place in private, however, it is possible that others may learn of an individual's study participation and, because of this, may treat them unfairly or discriminate against them.

## Phlebotomy

Participants may feel discomfort or pain when their blood is drawn. They may feel dizzy or faint or develop a bruise, swelling, small clot, or in rare cases, an infection where the needle goes into their arm.

#### Pelvic Examination and Procedures

Participants may feel discomfort, pain or pressure during the exam and when specimens are collected. They may have a small amount of vaginal bleeding or spotting which should stop shortly after the exam.

#### CVF Collection

Collection of CVF may cause discomfort or pressure in the vagina or genital area.

## Risks Associated with Vaginal Films

Participants may feel discomfort, itching, irritation, and vaginal discharge during film use. Based on previous film studies, these experiences are not prevalent.

#### Risks Associated with Placebo Excipients

All the excipients used in both films are generally regarded as safe (GRAS) and/or have a history of pharmaceutical use.

#### Social Harms

Although study sites will make every effort to protect participant privacy and confidentiality, it is possible that involvement in the study could become known to others and that social harms –

non-medical adverse consequences – may result. For example, participants could be treated unfairly, or could have problems being accepted by their families, partners and/or communities.

#### **13.4.2** Benefits

Participants in this study may experience no direct benefit. Participants and others may benefit in the future from information learned from this study. Specifically, information learned in this study may lead to the development of safe and effective interventions to prevent HIV acquisition and transmission. Participants also may appreciate the opportunity to contribute to the field of HIV prevention.

Participants will receive HIV/STI risk reduction counseling, HIV and STI testing, and physical and pelvic exams. Participants will be provided STI treatment free of charge, and referrals may be provided if needed. For other medical conditions identified as part of the study screening and/or follow-up procedures, participants will be referred to other sources of care available in their community. Some participants may have the opportunity to access expedient treatment and decreased morbidity due to early diagnosis and treatment of abnormalities identified during tests, examinations and referrals.

## **13.5 Informed Consent Process**

Written informed consent will be obtained from each study participant prior to screening. Written informed consent also will be obtained for long-term specimen storage and possible future testing, although consent for specimen storage is not required for study participation. In obtaining and documenting informed consent, the IoR and their designees will comply with applicable local and US regulatory requirements and will adhere to GCP and to the ethical principles that have their origin in the Declaration of Helsinki. Study staff must document the informed consent process in accordance with MATRIX's GDP guidelines (www.matrix4prevention.org). Participants will be provided with copies of the ICF if they are willing to receive them.

In addition to the ICF, the Protocol Team will work with study staff and community representatives to develop appropriate materials about the study and a standardized approach to the informed consent process to be implemented at study sites, which will be detailed in the MATRIX-002 SSP Manual.

The informed consent process will cover all elements of informed consent required by research regulations. In addition, the process specifically will address the following topics of importance to this study:

- The need to practice safer sex behaviors.
- Both study products are placebos that provide no protection against HIV acquisition, STIs, or pregnancy.
- The importance of adherence to the study visit and procedures schedule.
- The potential medical risks of study participation (and what to do if such risks are experienced).
- The potential social harms associated with study participation (and what to do if such harms are experienced).
- The limited benefits of study participation.

- The distinction between research and clinical care.
- The right to withdraw from the study at any time.

Furthermore, participants who agree to have their sexual partner contacted while in MATRIX-002 will be asked to read and sign an additional "Permission to Contact" form before the partner is invited to enroll. This form will explain that the participant gives the study staff permission to contact their sexual partner with the understanding that the partner will be invited to discuss their views on the film and its attributes and the participant's experiences using the vaginal film. This means the sexual partner will be aware of the participant's study involvement and use of the vaginal film. Sites will contact sexual partners according to site SOP and/or local IRB/IEC guidelines. Sexual partners who agree to enroll in the study will provide written informed consent prior to completing the IDI.

## 13.6 Participant Confidentiality

All study procedures will be conducted in private, and every effort will be made to protect participant privacy and confidentiality to the extent possible. Study sites will implement confidentiality protections that reflect the local study implementation plan and the input of study staff and community representatives to identify potential confidentiality issues and strategies to address them.

All study-related information will be stored securely at the study site. All participant information will be stored in locked areas with access limited to study staff. All laboratory specimens, study data collection, and administrative forms will be identified by coded participant number only to maintain participant confidentiality. All records that contain names or other personal identifiers, such as locator forms and ICFs, will be stored separately from study records identified by code number. All local databases will be secured with password protected access systems. Forms, lists, logbooks, appointment books, and any other listings that link participants' ID numbers to identifying information will be stored in a separate, locked file in an area with limited access. Participants' study information will not be released without their written permission, except as necessary for review, monitoring, and/or auditing by the following:

- Representatives of the US Federal Government, including the US OHRP, USAID, and/or contractors of USAID, and other local, US, or international regulatory authorities
- ACRO and ECS-HSR
- Representatives of Pitt/MWRIF
- MATRIX designees/representatives
- Study staff
- Site IRBs/IECs

## 13.7 Special Populations

## **13.7.1** Pregnant Women

Women who test positive for pregnancy at the Screening or Enrollment Visit will not be eligible to participate in this study. Should a participant test positive for pregnancy after Enrollment, a product discontinuation will be implemented. Follow-up visits and procedures will be discontinued, and the participant will be considered terminated from the study. An Early Termination Visit may

be completed and data collected per Section 7.4.2. During the informed consent process, participants will be informed that the placebo vaginal film is not a method of contraception and the effects of the placebo vaginal film on a developing human fetus are unknown.

#### 13.7.2 Children

The US NIH has mandated that children, defined as younger than 18 years old, be included in research trials when appropriate. This study meets "Justifications for Exclusion" criteria for younger children as set forth by the NIH (specifically, "insufficient data are available in adults to judge potential risk in children" and "children should not be the initial group to be involved in research studies"). As such, this study does not plan to enroll children.

## 13.8 Compensation

Pending IRB/IEC approval, participants will be compensated for time and effort in this study, and/or be reimbursed for travel to study visits and time away from work. Site-specific reimbursement amounts will be determined per local IRB/IEC/DRA guidelines and will be specified in the study ICFs of each individual site.

If a participant becomes ill or injured as a result of participation in this trial, medical treatment for the adverse reaction or injury will be provided appropriately. The site staff will refer the participant for ongoing treatment for the injury, if needed. Where required, clinical trial insurance purchased by sites will be responsible for compensating the study participant for appropriate medical expenses for treatment of any such illness or injury. An HIV infection that occurs during the course of the trial will not be considered an injury or illness caused by trial participation.

## 13.9 Reporting

## 13.9.1 Communicable Disease Reporting

Study staff will comply with local requirements to report communicable diseases including HIV identified among study participants to health authorities. Participants will be made aware of reporting requirements during the informed consent process.

## 13.9.2 Other Reporting

Study staff will comply with local requirements to report cases of sexual assault or of sexual activity involving a person below the age of consent identified in the study.

#### 13.10 Access to HIV-related Care

#### 13.10.1 HIV Counseling and Testing

HIV test-related counseling will be provided to all potential study participants who consent to undergo HIV screening to determine their eligibility for this study, and to all enrolled participants at each follow-up HIV testing time point. Testing will be performed in accordance with the algorithms in Appendix II. Counseling will be provided in accordance with standard HIV counseling policies and methods at each site and additionally will emphasize the unknown efficacy of the

study products in preventing HIV infection. Participants must receive their HIV test results to take part in this study. Condoms will be available to participants as part of standard risk reduction counseling.

## 13.10.2 Care for Participants Identified as HIV-Positive

An individual who has been identified as infected with HIV will be referred for management according to the local standard of care. Should a participant test positive for HIV after Enrollment Visit, follow-up procedures will be performed as per Section 7.4.1.

## 13.11 Study Discontinuation

This study may be discontinued at any time by USAID, MATRIX, Pitt/MWRIF, the OHRP, other local, US or international regulatory authorities, or site IRB/IEC.

## 14 PUBLICATION POLICY

USAID and MATRIX policies will govern publication of the results of this study. Any presentation, abstract, or manuscript will be submitted by the investigator to USAID, MATRIX and Pitt/MWRIF for review prior to submission.

## 15 APPENDICES

## **APPENDIX I: SCHEDULE OF STUDY VISITS AND EVALUATIONS**

| | | | | | | | _ | |
|---|---|---|---|---|---|---|---|---|
| | SCR<br>Visit 1 | Visit 2 (Day 0) | 24-72 hr<br>Contacts<br>Visits 3&7<br>(1-3 days<br>after V2&V6) | 1- & 2-wk<br>Contacts<br>Visits 4-5<br>(7&14 days<br>after V2) | 4-wk Visit<br>Visit 6<br>(28 days<br>after V2) | 6-wk<br>Contact<br>Visit 8<br>(14 days<br>after V6) | 8-wk<br>Visit<br>Visit 9<br>(28 days<br>after V6) | Final<br>Contact<br>Visit 10<br>(7 days<br>after V9) |
| ADMINISTRATIVE AND REGULATORY | | | | | | | | |
| Obtain/review informed consent for screening &/or enrollment (sites may split screening and enrollment consent if requested/required by IRB/IEC) | х | х | | | | | | |
| Assign a unique PTID | Х | | | | | | | |
| Collect demographic and background information | Х | | | | | | | |
| Assess/confirm eligibility | Х | Χ | | | | | | |
| Randomization | | Х | | | | | | |
| Confirm permission to contact sexual partner for IDI (subset) | | | | | | | х | |
| Collect/update/review contact/locator information | Х | Х | | Х | Х | Х | Х | Х |
| Provide reimbursement | Х | Х | X | Х | Χ | Х | Х | Х |
| Schedule next visit/contact | * | * | | Х | Χ | Х | Х | |
| COUNSELING | | | | | | l | | |
| HIV pre- and post-test counseling | Х | Х | | | Х | | Х | |
| HIV/STI risk reduction counseling | Х | Х | | | X | | Х | |
| Protocol counseling | Х | Χ | | * | Χ | * | Х | |
| BEHAVIORAL | | | | | | | | |
| Review instructional materials | | Х | | | Х | | | |
| Behavioral questionnaire(s) | | X<br>(pre & post<br>insertion) | | | Х | | Х | |
| Brief behavioral<br>assessment (concerns and<br>comfort with film use) | | | Х | Х | | Х | | |
| Social harms and benefits assessment | | | | | | | Х | |
| IDI – subset of participants | | | | | | | Хa | |
| IDI – sexual partners | | | | | | | Xp | |
| CLINICAL | | | | | | | | |
| Collect/update/review<br>medical and menstrual<br>history | Х | х | | Х | Х | Х | Х | Х |
| Collect/update/review concomitant medications | Х | Х | | Х | Х | Х | Х | Х |
| Physical exam (targeted after Screening) | Х | * | | | * | | * | |

| | | SCR<br>Visit 1 | ENR<br>Visit 2<br>(Day 0) | 24-72 hr<br>Contacts<br>Visits 3&7 | 1- & 2-wk<br>Contacts<br>Visits 4-5 | 4-wk Visit<br>Visit 6<br>(28 days | 6-wk<br>Contact<br>Visit 8 | 8-wk<br>Visit<br>Visit 9 | Final<br>Contact<br>Visit 10 |
|---|---|---|---|---|---|---|---|---|---|
| | | | | (1-3 days<br>after V2&V6) | (7&14 days<br>after V2) | after V2) | (14 days<br>after V6) | (28 days<br>after V6) | (7 days<br>after V9) |
| (ind | vic exam with speculum<br>cluding bimanual exam<br>Screening) | Х | Х | | | Х | | Х | |
| Visual examination by clinician to check vaginal film placement | | | Х | | | Х | | | |
| | n insertion assessment | | Х | | | Х | | | |
| | vide available test<br>ults | X | Х | | Х | Х | Х | X | Х |
| AE | assessment | | X | | X | X | X | X | Χ |
| | eat or prescribe<br>atment for RTI/UTI/STIs | * | * | | | * | | * | |
| | BORATORY | | | | | | ı | | |
| SALIVA | HIV test(s) (only at sites with CLIA certification) | Х | Х | | | Х | | х | |
| 뿔 | Urine pregnancy test | Χ | Χ | | | Χ | | X | |
| URINE | Urine dipstick/culture | * | * | | | * | | * | |
| | HIV test(s) (not<br>necessary for sites that<br>perform saliva testing) | X | Х | | | Х | | Х | |
| 8 | Plasma for archive | | Χ | | | | | | |
| ВГООБ | CBC | Χ | * | | | * | | Χ | |
| ш | Serum creatinine | Χ | * | | | * | | Χ | |
| | AST/ALT | Χ | * | | | * | | Χ | |
| | Syphilis serology | X | | | | | | | |
| | Pap test | ^ | | | | | | | |
| | KOH wet mount for candidiasis and/or BV | * | * | | | * | | * | |
| ELVIC | Vaginal Gram Stain | | Χ | | | Χ | | Х | |
| PEL | Vaginal swab(s) for microbiota | | Х | | | Х | | Х | |
| | Vaginal pH | | Χ | | | Χ | | Х | |
| | NAAT for GC/CT/TV | Х | Χ | | | Χ | | Х | |
| ST | UDY PRODUCT SUPPLY | | | | | | | | |
| | vide vaginal film for<br>f-insertion at clinic | | Х | | | Х | | | |
| Clir<br>film<br>par<br>atto | nician insertion of vaginal<br>n at clinic (only if<br>ticipant fails two<br>empts) | | Х | | | X | | V | |
| | er male condoms | | | | | Х | <u> </u> | X | |

X Required
\*If indicated and/or per local standard of care
^ if indicated (if participant is unable to provide documentation of a normal Pap test within 3 years prior to enrollment)
a At or after Visit 9, before Visit 10
b Within one month of participant Visit 9

## APPENDIX II: ALGORITHM FOR HIV TESTING – SCREENING/ENROLLING/FOLLOW-UP



\*CLIA certified labs may perform 1 rapid test

## APPENDIX III: SAMPLE INFORMED CONSENT FORM (SCREENING, ENROLLMENT, LONG-TERM STORAGE AND FUTURE TESTING)

#### SAMPLE INFORMED CONSENT FORM

# MATRIX-002 Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### **USAID**

Version 1.0 24 May 2023

**PRINCIPAL INVESTIGATOR:** [SITES TO INSERT]

**INSTITUTION:** [SITES TO INSERT]

**AFTER HOURS CONTACT DETAILS:** [SITES TO INSERT] **STUDY SITE CONTACT DETAILS:** [SITES TO INSERT]

**SHORT TITLE:** VALUE Placebo Film Study

## **INFORMED CONSENT**

[SITES TO INSERT APPROPRIATE GREETING] You are being invited to take part in this research study because you are an 18-45-year-old woman in good health. Approximately 100 women will take part in this study across sites in the United States (US), Kenya, South Africa, and Zimbabwe. This study is looking at two placebo vaginal films.

This study is sponsored by the US Agency for International Development (USAID) and conducted by the University of Pittsburgh/Magee-Womens Research Institute and Foundation (Pitt/MWRIF) as part of MATRIX: A USAID Project to Advance the Research and Development of Innovative HIV Prevention Products for Women. The placebo vaginal films are supplied by Pitt/MWRIF. At this site, the person in charge of this study is [SITES TO INSERT].

## **KEY INFORMATION**

- The study will assess the acceptability and safety of the two placebo vaginal films. The placebo films do not contain any active medication; the films do not prevent HIV.
- You would be randomly assigned to one of the two films and asked to use (self-insert) the
  assigned film two times (approximately one month apart). The study involves answering
  questions, undergoing pelvic examinations, and collecting blood and vaginal fluid samples.
- You would be in the study for approximately 9 weeks once you are enrolled.
- The study involves a total of 10 visits/contacts, including in person visits and telephone calls.
- There may be no benefit to participating.
- You cannot join this research study if you are living with HIV, pregnant, breastfeeding, or are already taking part in another research study involving drugs, medical devices, vaginal products, or vaccines.
- Taking part in this research study is voluntary. You do not have to participate, and you can stop your participation in the study at any time.

Please take the time to read this entire form and ask questions before deciding to join the study. If you are willing to take part in the study, you will sign this form. A copy of this form will be offered to you. Signing this form does not mean you will be able to join the study. You must first complete the screening tests and exams to see if you are eligible. It is important to know that your participation in this research study is your decision and taking part in this study is completely voluntary (see Your Rights as a Research Participant/Volunteer for more information).

## WHY IS THIS RESEARCH BEING DONE?

Investigators are studying products that women can use for HIV prevention. Vaginal films are being evaluated as one potential way to deliver anti-HIV drugs into the vagina (in future studies).

This study will allow participants to use one of the placebo vaginal films twice during their participation. The study will evaluate safety and will collect information on acceptability and use.

Both vaginal films being used in this study are 2 x 2 inch placebo vaginal films (contain no medication). They are "prototype" films for future studies and will be referred to as Film A and Film B. They differ by shape. The components of the placebo films being used in this study have been used in other products and/or have been generally regarded as safe.

#### WHO WILL BE IN THIS RESEARCH STUDY?

Approximately 100 women who are 18-45 years old will be enrolled in the study across sites in the United States (US), Kenya, South Africa, and Zimbabwe.

#### DO I HAVE TO BE IN THIS STUDY?

You do not have to be in this study. You can still get the care you need even if you do not join the study. If you join today, you can change your mind later.

## WHAT WILL I BE ASKED TO DO IF I JOIN THIS RESEARCH STUDY?

You will undergo a screening visit to be sure you are eligible and interested. If you are eligible and decide to enroll in this study, you will be asked to use (self-insert) one of two placebo vaginal films, approximately one month apart. Neither you nor investigators can choose the film you will use. Both placebo films are important to the study.

You must be using an effective method of birth control for at least two weeks before screening and agree to continue to use the method throughout the duration of the study to qualify.

At the Enrollment Visit (V2) you will be asked to insert the first vaginal film, undergo evaluations, and provide feedback about your experience. During the first month after film insertion, you will be asked to abstain from sex and not use anything in the vagina. For example, this means no sex, fingers, tampons, menstrual cups, toys, douches, vaginal medications. If you do not think you can agree to this, you should not participate.

Approximately a month later (V6) you will be asked to insert a second film (the same assigned film), undergo evaluations, and provide feedback about your experience. During the month following this 2<sup>nd</sup> film insertion, you will be permitted to have sex and use vaginal products if you choose.
You will have scheduled follow-up clinic visits and telephone contacts as detailed below.

# WHAT WILL HAPPEN DURING THE STUDY VISITS?

The study includes a total of ten (10) clinic visits or telephone contacts, including the Screening Visit today. All in-person visits will take place at this clinic. Telephone contacts may be done through a phone call or via text message. Participants who prefer to complete the telephone contacts in-person may elect to do so.

# **Study Visit Schedule:**



# **Screening Visit (Visit 1) Procedures:**

The procedures done at this visit will let us know if you can join this study and will take about [SITES TO SPECIFY TIMEFRAME].

At the Screening Visit, you will:

- Answer questions related to
  - o Demographics: date of birth, race, contact information, etc.
  - o Medical and menstrual history: review of any medical problems you may have
  - o Medication use: review any medication you take, including start date, dose, etc.
  - Birth control method: you must be using and agree to continue to use an acceptable, reliable method throughout the study to qualify
  - Visit questionnaire
- Undergo counseling
  - HIV/STI (sexually transmitted infection) counseling and how to reduce your risk
  - Abstinence (no sex and no vaginal product) counseling will be reviewed. This would be for the first month, starting at the Enrollment Visit.
    - It is important that you know if you are not currently using an acceptable method of contraception, or if you do not think you can abstain from vaginal intercourse or use of vaginal products for the first month of film use, you will not be eligible to participate in this study.

- Have examinations
  - Physical exam
  - Pelvic exam: a speculum (device inserted into the vagina) will be used to look at the vagina and cervix
- Have baseline testing:
  - o Urine pregnancy test: If you are pregnant, you will not be able to join
  - HIV test: [SITES TO INSERT TYPE OF HIV TEST and LOCAL REQUIRED LANGUAGE]
  - o Blood test: Approximately [SITES TO INSERT VOLUME] will be collected to look at the general health of your blood, basic kidney and liver function, and to screen for syphilis
  - o STI test for gonorrhea, chlamydia and trichomonas by collecting a Q-tip like swab
  - Pap smear: If you have not had a normal result within the required period and/or the report is not available, you will have a Pap smear performed by using a soft brush to collect a sample from your cervix [SITES TO MODIFY/ADD AS NEEDED: to screen for cervical cancer]
  - Additional tests may be done if you are having symptoms and as clinically indicated: urine dip stick/culture and/or microscope exam of vaginal fluid to check for infections
- Receive test results
  - Results of the tests listed above will be reviewed with you once available. Some tests results may be available while you are at today's visit (urine pregnancy test) while others may take up to a week to result (STI testing). The results of these tests will help to determine if you are eligible to participate.
  - If you are diagnosed with a urinary, vaginal (i.e., yeast or BV) or an STI at Screening, you will be offered/prescribed treatment
  - If there are other clinically significant findings, for example on your blood test or Pap smear, you will be referred for additional evaluations and treatment as needed
- In addition
  - Be provided reimbursement
  - May be tentatively scheduled for an Enrollment Visit within 45 days of Screening
    - Your menstrual cycle will be considered when scheduling your in-person visits because, ideally, no bleeding should occur around those visits

It may be necessary to conduct more than one clinic visit to complete all required screening procedures or if a test needs to be repeated.

If you do not join the study, blood and other samples collected at the Screening visit will not be kept or used for any tests other than those listed above.

If you are eligible and decide to enroll in the study, there are common study procedures that will happen at every in-person visit (V2, V6, V9), including:

- Review/update your contact information, including address and phone number\*
- Review/update your medical and menstrual history\*
- Review/update any medications you are taking/using\*
- Review/update any sexual activity or intravaginal product use
- Have HIV/STI testing and counseling [SITES TO MODIFY/ADD BELOW LANGUAGE AS NEEDED]
  - You will be told your test results as soon as they are available. You will talk with the study staff about the meaning of your results, how you feel about them, and learn about ways to prevent HIV and other STIs. Sometimes HIV tests are not

clearly positive, but also not clearly negative. In that case, we will do more tests until we are sure of your status. To participate in the study, you must receive the results of your HIV test. If the test shows you have HIV, you cannot join the study. We will refer you to available sources of medical care and other services you may need.

- Review of any new complaints or side effects once you start using the film\*
- Targeted physical exam, as clinically indicated based on symptoms/complaints
- Have a urine pregnancy test
- Have pelvic exam with collection of Q-tip swabs to look at the bacteria in the vagina
- As needed tests:
  - Repeat blood tests (general health of blood, kidney and liver function)
  - o Microscope exam of vaginal fluid to look for yeast or bacteria
  - Urine dip/culture
- Review of test results\*
- Treatment or referral for abnormal test results as needed
- Undergo protocol counseling, including HIV/STI risk reduction and contraceptive counseling, as needed\*
- Reimbursement for the study visit/contact\*
- Schedule next visit/contacts\*

# **Enrollment Visit (Visit 2) Procedures:**

Your Enrollment Visit (the visit where you enter the study) will take about [SITES TO SPECIFY TIMEFRAME]. You will be randomized to one of two vaginal placebo films at this visit. You will receive either placebo film A or B at this visit, to be self-inserted at the clinic.

The Enrollment Visit will take place up to 45 days after your Screening Visit.

In addition to the common study procedures listed above, at the Enrollment Visit, you will:

- Answer questions
  - About the vaginal film
  - About sexual behaviors and risk factors
  - Additional questions about the vaginal film following insertion
- Undergo counseling
  - o Abstinence (refrain from sex and vaginal products) counseling
- Have examinations
  - Pelvic exam prior to inserting film
  - Visual external (outside) genital exam after insertion of film to check placement
- Take a blood sample [SITES TO INSERT AMOUNT]. This blood sample will be stored in case there is a question about your test results at a later time.
- Be randomized to use Film A or B as described above
- Review instructional materials
  - You will be provided with vaginal film instruction materials to review prior to inserting the film. Study staff will be available to answer any questions you may have.
- Self-insert the assigned vaginal film (A or B)
  - o You will have two attempts to insert the vaginal film

<sup>\*</sup>These procedures will also be done at the scheduled Telephone Contacts (V4, V5, V8, V10)

 If after two attempts, you are having difficulty, a clinician will insert the film using a speculum

# 24-72-hour Phone Check-in (Visit 3) Procedures:

This contact will take place between 24-72 hours after insertion of the first film and will take approximately 5 minutes to complete.

You will be asked if you are having any issues or concerns with the film. You will be reimbursed for this contact.

# 1-week and 2-week Telephone Contacts (Visits 4 and 5) Procedures:

Your 1-week and 2-week follow-up contacts will take place approximately 7 and 14 days (one and two weeks) following the Enrollment Visit. These telephone contacts will take approximately [SITES TO SPECIFY TIMEFRAME] to complete.

In addition to the common study procedures with Telephone Contacts listed earlier, you will be asked about concerns and comfort with film use.

# 4-week Visit (Visit 6) Procedures:

This clinic visit will occur approximately 28 days (4 weeks) after the Enrollment Visit and will take between [SITES TO SPECIFY TIMEFRAME] to complete.

In addition to the common study procedures listed earlier, at this visit you will:

- Answer questions
  - About your experiences using the vaginal film
  - About sexual behaviors and use of vaginal products
  - o Additional questions about the vaginal film following insertion
- Undergo protocol instructions/counseling
  - o Reminder there are no restrictions on sex or vaginal product use
  - Explanation of (optional) sexual partner interview component
    - You will be given information to share with your partner to see if your partner would be comfortable participating in an interview
    - This is optional; if you don't feel comfortable including or asking your partner to participate, you will not be disqualified
    - Your partner would need to sign a separate consent
  - Offer male condoms
- Have examinations
  - o Pelvic exam with removal of any visible film from the first insertion
  - Visual external (outside) genital exam after insertion of second film to check placement
- Review instructional materials
  - You will be provided with vaginal film instruction materials to review prior to inserting the film. Study staff will be available to answer any questions you may have.
- Self-insert second vaginal film (A or B)
  - o You will be provided with your previously assigned vaginal film
  - o You will have two attempts to insert the vaginal film
  - If after two attempts, you are having difficulty, a clinician will insert the film using a speculum

# 24-72-hour Phone Check-in (Visit 7) Procedures:

This contact will take place between 24-72 hours after insertion of the second film and will take approximately 5 minutes to complete.

You will be asked if you are having any issues or concerns with the film. You will be reimbursed for this contact.

# 6-week Telephone Contact (Visit 8) Procedures:

Your 6-week follow-up contact will take place approximately 14 days (2 weeks) after Visit 6. This telephone contact will take between [SITES TO SPECIFY TIMEFRAME] to complete.

In addition to the common study procedures with Telephone Contacts listed earlier, you will be asked about concerns and comfort with film use.

# 8-week Visit (Visit 9) Procedures:

This clinic visit will occur approximately 28 days (4 weeks) after Visit 6 and will take between [SITES TO SPECIFY TIMEFRAME] to complete.

In addition to the common study procedures listed earlier, at this visit you will:

- Answer questions
  - About your experiences using the vaginal film
  - About sexual behaviors and use of vaginal products
  - o A subset of participants (up to 35 total) will be chosen to do an in-depth interview
    - If chosen, the interview will be performed [SITES TO SPECIFY MECHANISM: in the presence of one or two MATRIX-002 research staff members / remotely by a behavioral researcher]
    - Study staff will make every effort to ensure your privacy and confidentiality, and information you provide during the interview will not be shared with your partner
    - The interviewer may take notes, and interviews will be audio-recorded to make sure we record your words exactly how you said them
    - The interview will be focused on your experiences using the film and behaviors during the study and could take up to an hour to complete
    - The interview may occur during V9 or after up until V10
- Have examinations
  - o Pelvic exam and removal of any visible film
- Blood test: Approximately [SITES TO INSERT VOLUME] will be collected to look at the general health of your blood and basic kidney and liver function
- Offer male condoms
- In addition
  - Investigators will ask if you are willing to have your partner contacted to participate
    in an in-depth interview about your partner's experience while you were in the study.
    This is optional and you should only agree if you (and your partner) feel comfortable.
  - o If you agree, you will be asked to [SITES TO SPECIFY CONTACT METHOD: provide your partner's current contact information at this time / provide our contact information to your partner so they can call us if interested in participating]

# **Final Telephone Contact – Study Exit Visit (Visit 10) Procedures:**

Your Final Telephone Contact will take place approximately 7 days (one week) following Visit 9. This telephone contact will take approximately [SITES TO SPECIFY TIMEFRAME] to complete.

In addition to the common procedures with Telephone Contacts listed above, you will be asked about your wellness and any concerns. This will end your participation in the study.

#### **Additional Visits and Procedures**

In addition to the procedures listed above, it is possible that study clinicians may need to perform additional exams or tests, if necessary. For example, you may be asked to make additional clinic visits to perform these exams/tests if you report having symptoms and/or other issues, if there are abnormal test results, or due to mistakes during the collection, processing and/or shipping of your samples. These exams/tests might include the following:

- Physical and/or pelvic exam
- Test genital samples for STIs
- Test your urine for STIs or other infections
- Test your blood for STIs
- Test your blood to check the health of your blood, liver and kidneys
- Give you treatment or refer you for treatment of STIs or other issues, if needed.

It is important for you to complete every study visit/contact. If you cannot make a scheduled visit/contact, please tell the study staff as soon as possible so that the visit/contact can be rescheduled.

It is important that you remember that at any time during the study, study staff can answer any questions you may have about the procedures mentioned above or any other aspect of this study.

#### WHAT IF I BECOME INFECTED WITH HIV?

The placebo vaginal films do not contain medications and will not prevent HIV infection. Persons living with HIV will not be included in this study. Being in this study will not cause HIV infection. However, there is always a chance that you can get HIV through sex or other activities. If you become HIV-positive, you will stop using the study product and will stop taking part in this study. The study staff will refer you for medical care and other available services. The study does not pay for this care. [SITES TO INCLUDE/AMMEND THE FOLLOWING IF APPLICABLE: If you are interested, study staff will inform you of other available research studies you may be eligible for.]

Depending on local and national health requirements, the study staff may need to report certain diseases, including HIV. The reportable diseases at this site are [SITES TO INSERT]. We must inform the following [SITES TO INSERT MORE DETAILED INFORMATION REGARDING WHO WILL BE INFORMED OF THE REPORTABLE DISEASES]. [SITES TO INCLUDE/AMMEND THE FOLLOWING]: Outreach workers from the [LOCAL HEALTH AUTHORITY] may then contact you about informing your partner/s, since they also should be tested. If you do not want to inform your partner/s yourself, the outreach workers may contact them, according to the confidentiality quidelines of the [LOCAL HEALTH AUTHORITY].

# WHAT IF I BECOME PREGNANT?

The placebo vaginal films are not family planning methods and will not prevent pregnancy. We do not know what effect the study product(s) have on pregnancy, including any effect on the

unborn babies. Because of this, pregnant women may not join this study. Also, you must use an effective family planning method (e.g., birth control pills, hormonal-based methods, intrauterine device [IUD], the patch) other than a vaginal ring for at least two weeks before screening and for the study duration.

If you become pregnant during the study, study staff will refer you to available medical care and other services. The study does not pay for this care. You will stop using the study product and will stop taking part in this study. [SITES TO INCLUDE/AMMEND THE FOLLOWING IF APPLICABLE: If you are interested, study staff will inform you of other available research studies you may be eligible for.]

# **RISKS AND/OR DISCOMFORTS**

#### **Risks of Blood Draws**

You may feel discomfort or pain when your blood is drawn. You may feel dizzy or faint. You may have a bruise, swelling, small clot, or infection where the needle goes into your hand or arm.

#### **Risks of Pelvic Exams**

You may feel discomfort or pressure during the pelvic exam and collection of genital samples. You may have a small amount of vaginal bleeding or spotting which should stop shortly after the exam.

# **Risks of Vaginal Films**

You may feel discomfort, itching, irritation, and vaginal discharge during film use.

# **Risks of Placebo Excipients**

All the materials used in both films are generally regarded as safe and/or have a history of pharmaceutical use.

# Risks of HIV and Sexually Transmitted Infection (STI) Testing

HIV and STI testing may make you feel anxious regardless of the test results. Finding out your HIV status may also cause problems with your family, friends, or partner.

# **Other Possible Risks**

You may feel embarrassed and/or worried when talking about sexual activities (if you are currently sexually active), your living situation, ways to protect against HIV and STIs, and your test results. You can choose not to answer questions at any time. Trained study staff will help you with any feelings or questions you have.

We will make every effort to protect your privacy and confidentiality during the study visits. Your visits will take place in private. Reports via computer will be stored in computers that are password-protected and will not include personal information that could identify or link information to you; only your study ID number will be recorded. However, it is possible that others may learn of your participation in this study, and because of this, may treat you unfairly or discriminate against you. If you have any problems, study staff will talk with you and try to help you.

The in-depth interviews with study staff may be performed [SITES TO SPECIFY MECHANISM: at the clinic / remotely]. The interviews will be audio recorded and questions of a personal nature may be asked. Responding to these questions may make you uncomfortable. The audio files will be put into writing by the person conducting the interview or by another person who does not know you and does not have your personal information. You should NOT identify anyone in the interviews and any names that might be mentioned on the recording will only be noted in the transcript using a generic description. The audio files will be stored in computers that are password protected.

#### **BENEFITS**

Though you may not experience any direct benefit from participation in this study, information learned from this study may help us learn ways to prevent the spread of HIV in the future. Your opinions about the film are important to scientists working to develop this new prevention option. You will receive medical exams and counseling and testing for HIV and STIs. You will also have tests to check your overall health.

This study cannot give you general medical care, but study staff will refer you to another medical provider for care, if needed. Male condoms will be available at no cost, if you need them. If you are diagnosed with an STI during the study, you will receive medicine and/or a referral, if you need it.

# **NEW INFORMATION**

You will be told about any new information learned during this study that may affect your willingness to stay in the study. For example, we will let you know if we learn that the study product may be causing bad side-effects.

# WHY YOU MAY STOP USING THE STUDY PRODUCT EARLY OR BE ASKED TO LEAVE THE STUDY

You may need to leave the study early without your permission if:

- The study is cancelled by USAID, Pitt/MWRIF, the US Office for Human Research Protections (OHRP), MATRIX, the local government or regulatory agency, or the Institutional Review Board (IRB)/Independent Ethics Committee (IEC). An IRB/IEC is a committee that watches over the safety and rights of study participants.
- You are not able to keep appointments.
- Other reasons that may prevent you from completing the study successfully.

The study doctor will ask you to stop using the study products if:

- You acquire an HIV infection (see "If You Become Infected With HIV" section).
- You become pregnant or are breastfeeding (see "If You Become Pregnant" section).
- You use drugs for HIV prevention or to prevent infection after HIV exposure.
- You use injectable drugs for reasons other than treating disease.
- You experience a serious adverse event while on study.
- You fail to follow study requirements in a manner judged by the study doctor to significantly put you at risk of an adverse reaction or otherwise affect study outcomes.
- A study clinician decides that using the study product would be harmful to you, for example, you have a bad reaction to the vaginal film(s).

If a study doctor asks you to stop using study product, we will ask you to come in for an interim visit during which some/all of the procedures scheduled to occur on Visit 9 will be completed. You will then be exited from the study, unless otherwise informed by study staff.

#### **ALTERNATIVES TO BEING IN THE STUDY**

This is a placebo study enrolling healthy, adult women. You can choose not to participate in this study without affecting your care at this or other facilities or your ability to participate in other studies.

[SITES TO INCLUDE/AMEND THE FOLLOWING, IF APPLICABLE: You may be able to join other studies here or in the community. There may be other places where you can go for HIV counseling and testing and family planning. We will tell you about those studies and those places if you wish.]

# **COSTS TO YOU**

[SITES TO COMPLETE ACCORDING TO SITE CAPACITY] There is no cost to you for study visits, study products, physical/clinical exams, laboratory tests or other procedures. We can give you treatments for STIs (other than HIV) at no cost while you are in the study, or we can refer you for available treatment.

#### REIMBURSEMENT

[SITES TO INSERT INFORMATION ABOUT LOCAL REIMBURSEMENT:] You will receive [SITES TO INSERT AMOUNT \$XX] for your time, effort, and travel to and from the clinic for each scheduled study visit. You may receive [SITES TO INSERT AMOUNT \$XX] for any extra study visits. For responding to phone calls and text messages, you will receive up to [SITES TO INSERT AMOUNT \$XX]. If you are selected and agree to take part in the in-depth interview, you will receive [SITES TO INSERT AMOUNT \$XX].

# **CONFIDENTIALITY**

We will make every effort to keep your information private and confidential. But we cannot quarantee it.

Study visits will take place in private. We will keep the information about your study visits in a secure place that only certain people can access for the purposes of this study. We will only enter your information into computers protected by passwords and will not include information that could identify you. Your identity on these records will be indicated by a number rather than by your name, and the information linking these numbers with your name will be kept separate from the research records. You can choose not to answer questions at any time. We will keep the audio recordings and materials from all interviews and discussions confidential and will only use study numbers or fake names. We will store the original records, including the audio recordings, for at least three years after completion of the study. These records will be stored in a secure, locked location.

Your personal information may be disclosed if required by law. For example, if we learn something that would immediately put you or others in danger, the study staff must take steps to keep you and others safe. This means that we have to share any information with the authorities (hospital, police, or social services) that tells us you may be in danger. For example, if you tell us that you

plan to hurt or kill yourself, hurt or kill someone else, or if you tell us that someone is abusing or neglecting you.

The study staff may use your personal information to verify that you are not in any other research studies. This study will not use your name or identify you personally in any publication.

[SITES TO INSERT INFORMATION ABOUT SYSTEMS CURRENTLY IN PLACE TO ENSURE PARTICIPANTS ARE NOT PART OF OTHER CONFLICTING STUDIES, INCLUDING BIOMETRIC IDENTIFICATION SYSTEMS; SEE EXAMPLE BELOW FOR SOUTH AFRICAN SITES:

In clinical studies where study products or other medical devices are being assessed, it is important that volunteers are enrolled in only one clinical study at a time. Using more than one study product may lead to drug interactions and side effects that could potentially be harmful to your health. In addition to compromising the health of the study participant, this can affect the outcome of the study.

The Biometric Co-Enrollment Prevention System (BCEPS) is a web-based system developed by the South African Medical Research Council IT (Information Technology) department, for the prevention of co-enrolment (being enrolled in more than one study at a time). It is a secure system that is used to ensure participant safety and study integrity, in studies where co-enrolment could impact both.

Authorized study staff enters the South African Identify number (SA ID) or SA/foreign Passport Number of the participant into the system to check if they are enrolled in any study within any of the organizations using BCEPS in South Africa. During screening for a study at an Aurum Institute clinic/site, the SA ID number or SA/foreign Passport Number and all fingerprints are captured onto the system. At every study follow-up visit thereafter, their SA ID number or SA/foreign Passport Number and fingerprints will be checked.

In the long term, after study completion, it is important that study staff can verify what studies a participant has volunteered in, in order to ensure that the participant's safety is not compromised in future study participation. The SA ID number or SA/foreign Passport Number and fingerprints will remain in the database on an ongoing basis for a period of up to 15 years after the end of a study. If the participant has not participated in any additional studies for the 15-year period, their SA ID number or SA/foreign Passport Number and fingerprints will be removed from the system.

If a participant refuses for the system to be used at the initial visit or requests to be removed from the system while using a study product, the study investigator will decide if it is safe for the participant to be enrolled into the study or if it is safe to continue using study product without regularly checking for co-enrolment. The study that the potential participant is screening for may also prohibit co-enrolment in which case we will not be able to screen you.]

Your records may be reviewed by:

- Representatives of the US Federal Government, including US OHRP, USAID and/or USAID contractors, and other US, local or international regulatory authorities
- [SITES TO INSERT APPLICABLE LOCAL AND NATIONAL AUTHORITIES]
- Representatives of Pitt/MWRIF
- MATRIX representatives

- Study monitors
- Site IRB/IEC
- Study staff

[US SITE TO INCLUDE/AMEND THE FOLLOWING: Federal and state laws and the federal medical Privacy Rule also protect your privacy. By signing this form, you provide your authorization for the use and disclosure of information protected by the Health Insurance Portability and Accountability Act (HIPAA) Privacy Rule. This includes things learned from the procedures described in this consent form. Study staff may also collect other information including your name, address, date of birth, and information from your medical records.]

[NON-US SITES TO INCLUDE/AMEND THE FOLLOWING: As part of your participation in this research study, your personal information may be sent to the United States for analysis or storage. This includes things learned from the procedures described in this consent form. Study staff may also collect other information including your name, address, date of birth, and information from your medical records. There are laws in the U.S. to protect your personal information when in that country.]

[SOUTH AFRICA SITES TO INCLUDE/AMEND THE FOLLOWING: The Protection of Personal Information Act (POPIA) ensures that all South African institutions collect, process, store, and share your personal information in a responsible manner and that they will be held accountable should they abuse or compromise your personal information.]

People outside the study team may need to see or receive your information for this study, such as those listed above. We cannot do this study without your authorization to use and give out your information to them. You do not have to give us this authorization. If you do not, then you may not join this study.

The use and disclosure of your information has no time limit. You may cancel your authorization to use and disclose your information at any time by notifying the Principal Investigator of this study in writing. If you do cancel your authorization to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study, or information we disclosed before you wrote to the Principal Investigator to cancel your authorization.

# **RESEARCH-RELATED INJURY**

[SITES TO INCLUDE/AMMEND PER THEIR INSTITUTIONAL POLICY: It is unlikely that you will be injured by being in this study. If you are injured or get sick from being in this study, please tell study staff immediately.

If you believe that the research procedures have resulted in an injury to you, immediately contact the Principal Investigator who is listed on the first page of this form. If you become ill or injured as a result of participation in this study, medical treatment for the adverse reaction or injury will be provided appropriately. The site staff will refer you for ongoing treatment for the injury, if needed. Clinical trial insurance purchased by the site will be responsible for compensating you for appropriate medical expenses for treatment of any such illness or injury. An HIV infection that occurs during the course of the trial will not be considered an injury or illness caused by trial

participation. The research center or sponsor is not responsible for any loss, injuries and/or damages that are caused by any of the following things:

- Any injury that happens because you used other medicine during the study that you did not tell us about.
- Any injury that happens because you did not follow instructions given by the study doctor or nurse.
- Any injury that happens because of negligence on your part.]

SITES TO SPECIFY ANY ADDITIONAL POLICY RELATED TO EMERGENCY MEDICAL ATTENTION

[US SITE TO INCLUDE/AMEND THE FOLLOWING: To pay these medical expenses, Pitt/MWRIF will need to know some information about you, like your name, date of birth, and social security number or Medicare Health Insurance Claim Number. This is because they have to check to see if you receive Medicare and if you do, report the payment it makes to Medicare.]

You are not giving up any legal rights by signing this form.

# **CLINICALTRIALS.GOV**

A description of this research study will be available on https://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

[SOUTH AFRICA SITES TO INCLUDE LANGUAGE RELATED TO SOUTH AFRICAN NATIONAL CLINICAL TRIALS REGISTER]

#### YOUR RIGHTS AS A RESEARCH PARTICIPANT/VOLUNTEER

[SITES TO SPECIFY INSTITUTIONAL POLICY:] Being in this study is completely voluntary. You may choose not to join this study or leave this study at any time. If you choose not to join or to leave the study, you can still join other studies and you can still access non-study services you would normally get at this or another clinic. If you leave the study, your specimens will be destroyed when all protocol-specified testing has been completed and your study records may be kept for at least three years after study completion. If you want the results of the study after it is over, let the study staff members know.

# **PROBLEMS OR QUESTIONS**

If you ever have any questions about the study, or if you have a research-related injury, you should contact [INSERT NAME OF THE INVESTIGATOR OR OTHER STUDY STAFF] at [INSERT TELEPHONE NUMBER AND/OR PHYSICAL ADDRESS].

If you have questions about your rights as a research participant, you should contact [INSERT NAME OR TITLE OF PERSON ON THE IRB/EC OR OTHER ORGANIZATION APPROPRIATE FOR THE SITE] at [INSERT PHYSICAL ADDRESS AND TELEPHONE NUMBER].

[SITES TO OMIT THE FOLLOWING IF A SEPARATE CONSENT FOR STORAGE AND FUTURE TESTING OF SPECIMENS IS REQUIRED]

# CONSENT FOR LONG-TERM STORAGE AND FUTURE TESTING OF SPECIMENS and RELATED HEALTH INFORMATION

There might be a small amount of blood or genital samples left over after we have done all of the study-related testing. We would like to ask your permission to store these leftover samples and related health information for use in future studies, such as future research to fight HIV and other related diseases. This health information may include personal facts about you such as your race, ethnicity, sex, medical conditions and your age range. This health information will not include your name or any personal identifying information. The samples will be stored by your participant number only.

If you enroll in the study and agree, your samples and related health data will be stored safely and securely at facilities that are designed so that only approved researchers will have access to the samples. Some employees of the facilities will need to have access to your samples to store them and keep track of where they are, but these people will not have information that directly identifies you.

There is no time limit on how long your samples will be stored. Your samples may be shipped and/or stored outside of the country. The type of testing planned for your leftover specimens is not yet known. However, samples may be used by Pitt/MWRIF to complete additional quality assurance testing, ensuring that the tests work correctly and supply accurate data. No genetic testing on either a limited set or the full set of genes is planned for leftover samples that are stored for the purposes of future research. It is important that you know that any future testing or studies planned for these specimens must be approved by an Institutional Review Board before they can be done. You will not receive the results from any future testing of these specimens.

You can still enroll in this study if you decide not to have leftover samples stored for future studies. If you do not want the leftover samples stored, we will destroy them when all protocol-specified testing has been completed. You can withdraw your consent for the storage and future testing of specimens at any time by providing your request in writing to the person in charge of this study. However, researchers will not be able to destroy samples or information from research that is already underway.

| Initials and Date | I DO agree to allow my biological specimens and health data to be stored and used in future research studies. I understand my biological specimens may be shipped and stored outside of the country. |
|---|---|
| Initials and Date | I DO NOT agree to allow my biological specimens and health data to be stored and used in future research studies. |

[SITES TO OMIT THE FOLLOWING IF A SEPARATE CONSENT IS REQUIRED FOR PARTICIPANT IDI]

#### **CONSENT TO PARTICIPATE IN AN IN-DEPTH INTERVIEW**

We would like to ask your permission to participate in a conversation-style interview (in-depth interview or IDI) at the end of the study to gather more feedback about the placebo vaginal film. If you agree and are selected to participate in the IDI, trained study staff will ask you questions about your experiences using the product, about product design, packaging and delivery, and other topics related to product use. Information you provide during the IDI will not be shared with your partner. The IDI may be conducted at the study site, over a secure digital platform, or an agreed upon location.

The IDI is anticipated to last approximately 45-60 minutes. Study staff will take notes and record the interview. You can choose not to answer questions at any time. We will keep the audio recordings and materials from all interviews and discussions confidential and will only use study numbers or fake names to identify them. These materials will be stored in a secure, locked location for at least three years after completion of the study.

We will reconfirm the decision you make today at later study visits should you change your mind about participating in the IDI.

You can still enroll in this study if you decide not to participate in the IDI. You can withdraw your consent to participate in the IDI at any time.

| Initials and Date | I DO agree to participate in an in-depth interview. I understand the interview will be recorded and notes will be taken. |
|---|---|
| <br>Initials and Date | I DO NOT agree to participate in an in-depth interview. |

[SITES TO OMIT THE FOLLOWING IF A SEPARATE CONSENT IS REQUIRED FOR PERMISSION TO CONTACT SEXUAL PARTNER]

# PERMISSION TO CONTACT SEXUAL PARTNER

We would like to ask your permission to contact your sexual partner to participate in a conversation-style interview (in-depth interview or IDI) at the end of the study to gather more feedback about the vaginal film.

If both of you agree and your partner is selected to participate in the IDI, trained study staff will ask your partner questions about their views on the vaginal film and its characteristics and about your experiences using the vaginal film. This means that your partner will be aware of your participation in this study and your use of the vaginal film but no other information will be shared with your partner.

If you give us permission to talk to your sexual partner, you will be asked to [SITES TO SPECIFY CONTACT METHOD: provide their current contact information at this time / provide our contact information to your partner so they can call us if interested in participating].

We will reconfirm the decision you make today at later study visits should you change your mind about us contacting your sexual partner.

You can still enroll in this study if you decide not to give us permission to contact your sexual partner. You can withdraw your permission for us to contact your sexual partner at any time.

| Initials and Date | I DO give permission for study staff to talk to my sexual partner. I agree to [SITES TO SPECIFY CONTACT METHOD: provide current contact information for my sexual partner / provide my partner with your contact information so they can call you for more information]. |
|---|---|
| Initials and Date | I DO NOT give permission for study staff to talk to my sexual partner. |

# [SITES TO OMIT THE FOLLOWING IF NOT APPLICABLE]

# **CONSENT FOR OFF-SITE VISITS**

If the site determines that an off-site visit is appropriate and with your permission, members of the research team at this clinic may be able to schedule off-site visits with you at your home or at another location as part of the study. Some of the scheduled study visits and some of the study procedures may take place at your home or other location outside of the research clinic. For example, if you need to receive study product or to have a urine or blood sample collected but you are unable to come into the clinic. The study personnel will explain in greater detail the requirements of these visits (like the conditions of the place, the type of visit and the time it will take) and the procedures in-place to maintain your information in a confidential manner. However, it is important that you know that off-site visits may eventually affect your confidentiality even if the study staff take precautions not to disclose the purpose of the visits.

We will only conduct visits outside of the clinic if you give us permission to do so. Please read carefully the following statement and initial and date one option. Choosing not to have study visit procedures outside of the study clinic will not affect your participation in this study. Even if you agree today, you can withdraw your consent for off-site visits at any time by providing your request in writing to the person in charge of this study. In addition, before each off-site visit, we will confirm with you that you still agree and remember today's discussion.

| PARTICIPANT INITIALS | | |
|---|---|---|
| Initials | Date | I DO agree to have study visit procedures at a location other than the study clinic by clinic staff, when necessary. |
| Initials | Date | I DO NOT agree to have study visit procedures at a location other than the study clinic by clinic staff, when necessary. |

#### SIGNATURE PAGE

[INSERT SIGNATURE BLOCKS AS REQUIRED BY THE LOCAL IRB/IEC:]

All of the above has been explained to me and all of my current questions have been answered. I understand that I can ask questions about any aspect of this research study during the course of this study, and that future questions will be answered by the researchers listed on the first page of this form or their representatives.

Any questions I have about my rights as a research participant will be answered by [INSERT LOCAL IRB/IEC INFORMATION].

I voluntarily agree to be in this research study. A copy of this permission form will be given to me.

| Participant's Name (Print) | _ |
|-------------------------------------------------------------|------|
| Participant's Signature | Date |
| Study Staff's Name Conducting<br>Consent Discussion (Print) | |
| Study Staff Conducting<br>Consent Discussion (Signature) | Date |
| Witness Name (Print) | _ |
| Witness Signature | Date |

# APPENDIX IV: SAMPLE INFORMED CONSENT FORM (SEXUAL PARTNER SUBSET)

#### SAMPLE INFORMED CONSENT FORM

# MATRIX-002 Trial to Assess Acceptability and Safety of Two Placebo Prototype Vaginal Films

#### **USAID**

Version 1.0 24 May 2023

**PRINCIPAL INVESTIGATOR:** [SITES TO INSERT]

**INSTITUTION:** [SITES TO INSERT]

**AFTER HOURS CONTACT DETAILS:** [SITES TO INSERT] **STUDY SITE CONTACT DETAILS:** [SITES TO INSERT]

**SHORT TITLE:** VALUE Placebo Film Study

# **INFORMED CONSENT**

[SITES TO INSERT APPROPRIATE GREETING] You are being invited to take part in this research study because you were identified by a MATRIX-002 study participant as their sexual partner. MATRIX-002 is looking at two placebo vaginal films. Up to 30 sexual partners of MATRIX-002 participants like you will take part in this study across sites in the United States (US), Kenya, South Africa, and Zimbabwe.

This study is sponsored by the US Agency for International Development (USAID) and conducted by the University of Pittsburgh/Magee-Womens Research Institute and Foundation (Pitt/MWRIF) as part of MATRIX: A USAID Project to Advance the Research and Development of Innovative HIV Prevention Products for Women. At this site, the person in charge of this study is [SITES TO INSERT].

#### **KEY INFORMATION**

- There are no study products (investigational drugs or other products) for you to use in this research study.
- The purpose of including sexual partners in this study is to better understand your views about the vaginal film and its characteristics, and your views on your partner's experiences using the vaginal film.
- If you qualify and choose to participate, you will be enrolled in the study and asked to complete one conversation-style interview (in-depth interview) with trained study staff. The total length of your participation in the study will be one visit of approximately [SITES TO SPECIFY TIMEFRAME].
- Some risks or discomforts from participating in this study include:
  - Feeling uncomfortable with some of the questions study staff may ask about your sexual behaviors and relationships.

- Risk of conflict in your relationship if you or your partner are upset by discussions of sex, contraceptive choice, or HIV prevention.
- There may be no benefit to participating.
- Taking part in this research study is voluntary. You do not have to participate, and you can stop your participation in the study at any time.

Please take the time to read this entire form and ask questions before deciding to join the study. If you are willing to take part in the study, you will sign this form. A copy of this form will be offered to you. Signing this form does not mean you will be able to join the study. You must first complete the screening assessment to see if you are eligible. It is important to know that your participation in this research study is your decision and taking part in this study is completely voluntary (see Your Rights as a Research Participant/Volunteer for more information).

#### WHY IS THIS RESEARCH BEING DONE?

Investigators are studying products that women can use for HIV prevention. Vaginal films are being evaluated as one potential way to deliver anti-HIV drugs into the vagina (in future studies). The MATRIX-002 study involves two placebo vaginal films (containing no medication). The components of both placebo films used in this study have been used in other products and/or have been generally regarded as safe.

The main goal of including sexual partners like you in this study is to better understand your views about the vaginal film and its characteristics, and your views on your partner's experiences using the vaginal film during the study.

# WHO WILL BE IN THIS RESEARCH STUDY?

Up to 30 sexual partners of MATRIX-002 participants will be enrolled in the study across various sites in the United States (US), Kenya, South Africa, and Zimbabwe.

# DO I HAVE TO BE IN THIS STUDY?

You do not have to be in this study. You can still get the care you need even if you do not join the study.

# WHAT WILL I BE ASKED TO DO IF I JOIN THIS RESEARCH STUDY?

You will be asked to participate in an in-depth interview (IDI) with trained study staff. You will be asked about your attitudes towards and experiences with the vaginal film, and your perspective of your partner's attitudes and experiences with the vaginal film.

# WHAT WILL HAPPEN DURING THE STUDY VISIT?

The study consists of one study visit, which will take place after you sign this informed consent form. If you agree and are eligible to participate, the IDI may take place today. If scheduling does not allow, it may take place on a different day that is convenient for you. Additional visit(s) may be conducted to complete all required procedures, if necessary. The visit will take place at a place agreed upon by you and the study staff, which may be the study clinic, your home, or another convenient location [SITE TO INCLUDE ALTERNATE LOCATION].

The procedures done at this visit will take about [SITES TO SPECIFY TIMEFRAME].

• Study staff will ask you where you live and other questions about you, and your understanding of the study requirements.

- In the IDI, you will be asked questions about:
  - o Your age, education level, health, relationship status, and employment status.
  - Your views about HIV risk and prevention, sexual history, existing prevention methods, and aspects of your relationship.
  - Your views about the vaginal film and your partner's experiences using the vaginal film
- The IDI will be performed [SITES TO SPECIFY MECHANISM: in the presence of one or two MATRIX-002 research staff members / remotely by a behavioral researcher]. The IDI will take approximately [SITES TO SPECIFY TIMEFRAME].
  - Study staff will make every effort to ensure your privacy and confidentiality. Information you provide during the IDI will not be shared with your partner.
  - During the IDI, the interviewer may take notes. Interviews will be audio-recorded to make sure we record your words exactly how you said them.
- In addition, study staff will:
  - Reimburse you for your visit.
  - o Inform you about other available health and social services, if needed.
  - Schedule your next visit, if necessary.

# **RISKS AND/OR DISCOMFORTS**

You may feel embarrassed and/or worried when talking about sexual activities, your living situation, or your opinions about HIV prevention strategies. You can choose not to answer questions at any time. Trained study staff will help you with any feelings or questions you have.

We will make every effort to protect your privacy and confidentiality during the study visit. Your visit will take place in private. Reports via computer will be stored in computers that are password-protected and will not include personal information that could identify or link information to you; only your study ID number will be recorded. However, it is possible that others may learn of your participation in this study, and because of this, may treat you unfairly or discriminate against you. If you have any problems, study staff will talk with you and try to help you.

The interviews with study staff will be audio recorded and questions of a personal nature may be asked. Responding to these questions may make you uncomfortable. The audio files will be put into writing by the person conducting the interview or by another person who does not know you and does not have your personal information. You should NOT identify anyone in the interviews and any names that might be mentioned on the recording will only be noted in the transcript using a generic description. The audio files will be stored in computers that are password protected.

#### **BENEFITS**

Though you may not experience any direct benefit from participation in this study, information learned from this study may help us learn ways to prevent the spread of HIV in the future. Your opinions about the film are important to scientists working to develop this new prevention option.

Medical care for HIV infection and other health conditions will not be part of this study. This study cannot provide you with general medical care, but study staff will refer you to other available sources of care, if needed.

#### **NEW INFORMATION**

You will be told when study results may be available, and how to learn about them.

#### **COSTS TO YOU**

There is no cost to you for study-related visits.

#### REIMBURSEMENT

[SITES TO INSERT INFORMATION ABOUT LOCAL REIMBURSEMENT:] You will receive [SITES TO INSERT AMOUNT \$XX] for your time, effort, and travel to and from the clinic to take part in the in-depth interview.

#### **CONFIDENTIALITY**

We will make every effort to keep your information private and confidential. But we cannot guarantee it.

The study visit will take place in private. We will keep the information about your study visit in a secure place that only certain people can access for the purposes of this study. We will only enter your information into computers protected by passwords and will not include information that could identify you. Your identity on these records will be indicated by a number rather than by your name, and the information linking these numbers with your name will be kept separate from the research records. You can choose not to answer questions at any time. We will keep the audio recordings and materials from all interviews and discussions confidential and will only use study numbers or fake names. We will store the original records, including the audio recordings, for at least three years after completion of the study. These records will be stored in a secure, locked location.

Your personal information may be disclosed if required by law. For example, if we learn something that would immediately put you or others in danger, the study staff must take steps to keep you and others safe. This means that we have to share any information with the authorities (hospital, police, or social services) that tells us you may be in danger. For example, if you tell us that you plan to hurt or kill yourself, hurt or kill someone else, or if you tell us that someone is abusing or neglecting you.

This study will not use your name or identify you personally in any publication.

Your records may be reviewed by:

- Representatives of the US Federal Government, including US OHRP, USAID and/or USAID contractors, and other US, local or international regulatory authorities
- [SITES TO INSERT APPLICABLE LOCAL AND NATIONAL AUTHORITIES]
- Representatives of Pitt/MWRIF
- MATRIX representatives
- Study monitors
- Site IRB/IEC
- Study staff

[US SITE TO INCLUDE/AMEND THE FOLLOWING: Federal and state laws and the federal medical Privacy Rule also protect your privacy. By signing this form, you provide your authorization for the use and disclosure of information protected by the Health Insurance Portability and

Accountability Act (HIPAA) Privacy Rule. This includes things learned from the procedures described in this consent form. Study staff may also collect other information including your name, address, date of birth, and information from your medical records.]

[NON-US SITES TO INCLUDE/AMEND THE FOLLOWING: As part of your participation in this research study, your personal information may be sent to the United States for analysis or storage. This includes things learned from the procedures described in this consent form. Study staff may also collect other information including your name, address, date of birth, and information from your medical records. There are laws in the U.S. to protect your personal information when in that country.]

[SOUTH AFRICA SITES TO INCLUDE/AMEND THE FOLLOWING: The Protection of Personal Information Act (POPIA) ensures that all South African institutions collect, process, store, and share your personal information in a responsible manner and that they will be held accountable should they abuse or compromise your personal information.]

People outside the study team may need to see or receive your information for this study, such as those listed above. We cannot do this study without your authorization to use and give out your information to them. You do not have to give us this authorization. If you do not, then you may not join this study.

The use and disclosure of your information has no time limit. You may cancel your authorization to use and disclose your information at any time by notifying the Principal Investigator of this study in writing. If you do cancel your authorization to use and disclose your information, your part in this study will end and no further information about you will be collected. Your cancellation would not affect information already collected in the study, or information we disclosed before you wrote to the Principal Investigator to cancel your authorization.

# **RESEARCH-RELATED INJURY**

[SITES TO INCLUDE/AMMEND PER THEIR INSTITUTIONAL POLICY: It is unlikely that you will be injured by being in this study. If you are injured or get sick from being in this study, please tell study staff immediately.

If you believe that the research procedures have resulted in an injury to you, immediately contact the Principal Investigator who is listed on the first page of this form. If you become ill or injured as a result of participation in this study, medical treatment for the adverse reaction or injury will be provided appropriately. The site staff will refer you for ongoing treatment for the injury, if needed. Clinical trial insurance purchased by the site will be responsible for compensating you for appropriate medical expenses for treatment of any such illness or injury. An HIV infection that occurs during the course of the trial will not be considered an injury or illness caused by trial participation. The research center or sponsor is not responsible for any loss, injuries and/or damages that are caused by any of the following things:

- Any injury that happens because you used other medicine during the study that you did not tell us about.
- Any injury that happens because you did not follow instructions given by the study doctor or nurse.
- Any injury that happens because of negligence on your part.

SITES TO SPECIFY ANY ADDITIONAL POLICY RELATED TO EMERGENCY MEDICAL ATTENTION

[US SITE TO INCLUDE/AMEND THE FOLLOWING: To pay these medical expenses, Pitt/MWRIF will need to know some information about you, like your name, date of birth, and social security number or Medicare Health Insurance Claim Number. This is because they have to check to see if you receive Medicare and if you do, report the payment it makes to Medicare.]

You are not giving up any legal rights by signing this form.

#### **CLINICALTRIALS.GOV**

A description of this research study will be available on https://www.ClinicalTrials.gov, as required by U.S. law. This website will not include information that can identify you. At most, the website will include a summary of the results. You can search this website at any time.

[SOUTH AFRICA SITES TO INCLUDE LANGUAGE RELATED TO SOUTH AFRICAN NATIONAL CLINICAL TRIALS REGISTER]

# YOUR RIGHTS AS A RESEARCH PARTICIPANT/VOLUNTEER

[SITES TO SPECIFY INSTITUTIONAL POLICY:] Being in this study is completely voluntary. You may choose not to join this study or leave this study at any time. If you choose not to join or to leave the study, you can still join other studies and you can still access non-study services you would normally get at this clinic. If you leave the study, your study records may be kept for at least three years after study completion. If you want the results of the study after it is over, let the study staff members know.

# **PROBLEMS OR QUESTIONS**

If you ever have any questions about the study, or if you have a research-related injury, you should contact [INSERT NAME OF THE INVESTIGATOR OR OTHER STUDY STAFF] at [INSERT TELEPHONE NUMBER AND/OR PHYSICAL ADDRESS].

If you have questions about your rights as a research participant, you should contact [INSERT NAME OR TITLE OF PERSON ON THE IRB/EC OR OTHER ORGANIZATION APPROPRIATE FOR THE SITE] at [INSERT PHYSICAL ADDRESS AND TELEPHONE NUMBER].

#### SIGNATURE PAGE

[INSERT SIGNATURE BLOCKS AS REQUIRED BY THE LOCAL IRB/IEC:]

All of the above has been explained to me and all of my current questions have been answered. I understand that I can ask questions about any aspect of this research study during the course of this study, and that future questions will be answered by the researchers listed on the first page of this form or their representatives.

Any questions I have about my rights as a research participant will be answered by [INSERT LOCAL IRB/IEC INFORMATION].

I voluntarily agree to be in this research study. A copy of this permission form will be given to me.

| Participant's Name (Print) | _ |
|-------------------------------------------------------------|----------|
| Participant's Signature | Date |
| Study Staff's Name Conducting<br>Consent Discussion (Print) | |
| Study Staff Conducting<br>Consent Discussion (Signature) | <br>Date |
| Witness Name (Print) | |
| Witness Signature | <br>Date |

#### REFERENCES

- Alternative Formulations of Tenofovir and UC781. <a href="https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/8471636">https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/8471636</a>.
   <a href="https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/8471636">https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/8471636</a>.
   <a href="https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/8471636">https://reporter.nih.gov/search/K5gvxVFx3ECPmIAo3Bt15Q/project-details/84716
- Film Antiretroviral Microbicide Evaluation. <a href="https://reporter.nih.gov/search/HcBIzL\_XW0SbUQ2QIZ5krA/project-details/9707725">https://reporter.nih.gov/search/HcBIzL\_XW0SbUQ2QIZ5krA/project-details/9707725</a>, February 23, 2023.
- Acceptability Study of Vaginal Films for HIV Prevention (FACE). <a href="https://clinicaltrials.gov/ct2/show/NCT01231763?term=NCT01231763&draw=2&rank=1">https://clinicaltrials.gov/ct2/show/NCT01231763?term=NCT01231763&draw=2&rank=1</a>. Accessed February 23, 2023.
- 4. Patel SK, Bunge K, Downs J, Hillier S, Rohan L. Vaginal Film Administration and Placement Study in Women (FLAG Trial). Paper presented at: Aids Research and Human Retroviruses2018.
- 5. Musara P, Milford C, Shapley-Quinn MK, et al. Preferences and Acceptability of Vaginal Delivery Forms for HIV Prevention Among Women, Male Partners and Key Informants in South Africa and Zimbabwe: Qualitative Findings. *AIDS Behav.* Jan 2021;25(1):124-138.
- 6. Nel AM, Mitchnick LB, Risha P, Muungo LT, Norick PM. Acceptability of vaginal film, soft-gel capsule, and tablet as potential microbicide delivery methods among African women. *J Womens Health (Larchmt).* Aug 2011;20(8):1207-1214.
- 7. Guthrie KM, Fava JL, Vargas SE, et al. The Role of Volume in the Perceptibility of Topical Vaginal Formulations: User Sensory Perceptions and Experiences of Heterosexual Couples During Vaginal Sex. *AIDS Res Hum Retroviruses.* Dec 2020;36(12):1059-1070.
- 8. Guthrie KM, Rohan L, Rosen RK, et al. Vaginal film for prevention of HIV: using visual and tactile evaluations among potential users to inform product design. *Pharm Dev Technol.* Mar 2018;23(3):311-314.
- 9. Bunge KE, Dezzutti CS, Rohan LC, et al. A Phase 1 Trial to Assess the Safety, Acceptability, Pharmacokinetics, and Pharmacodynamics of a Novel Dapivirine Vaginal Film. *J Acquir Immune Defic Syndr*. Apr 15 2016;71(5):498-505.
- 10. Robinson JA, Marzinke MA, Bakshi RP, et al. Comparison of Dapivirine Vaginal Gel and Film Formulation Pharmacokinetics and Pharmacodynamics (FAME 02B). *AIDS Res Hum Retroviruses*. Apr 2017;33(4):339-346.
- 11. Politch JA, Cu-Uvin S, Moench TR, et al. Safety, acceptability, and pharmacokinetics of a monoclonal antibody-based vaginal multipurpose prevention film (MB66): A Phase I randomized trial. *PLoS Med.* Feb 2021;18(2):e1003495.
- 12. Bunge KE, Dezzutti CS, Hendrix CW, et al. FAME-04: A Phase 1 trial to assess the safety, acceptability, pharmacokinetics and pharmacodynamics of film and gel formulations of tenofovir. *J Int AIDS Soc.* Aug 2018;21(8):e25156.
- 13. Robinson JA, Marzinke MA, Fuchs EJ, et al. Comparison of the Pharmacokinetics and Pharmacodynamics of Single-Dose Tenofovir Vaginal Film and Gel Formulation (FAME 05). *J Acquir Immune Defic Syndr*. Feb 1 2018;77(2):175-182.
- 14. A Study of the Safety and Acceptability of a Placebo Vaginal Film: FAME101 (FAME101). <a href="https://clinicaltrials.gov/ct2/show/NCT03537092?term=NCT03537092&draw=2&rank=1">https://clinicaltrials.gov/ct2/show/NCT03537092?term=NCT03537092&draw=2&rank=1</a>. Accessed February 23, 2023.
- 15. Safety and Pharmacokinetics of Two Vaginal Film Formulations Containing the Integrase Inhibitor MK-2048 (FAME103).

- https://clinicaltrials.gov/ct2/show/NCT04319718?term=NCT04319718&draw=2&rank=1. Accessed February 23, 2023.
- 16. Randomized Cross-Over Study of Self-Insertion of Two Placebo Vaginal Film Formulations (FAME103B). <a href="https://clinicaltrials.gov/ct2/show/NCT04391036?term=NCT04391036&draw=2&rank=1">https://clinicaltrials.gov/ct2/show/NCT04391036?term=NCT04391036&draw=2&rank=1</a>. Accessed February 23, 2023.
- 17. Long Acting Film Technology for Contraception and HIV Prevention (LATCH). <a href="https://reporter.nih.gov/search/qr4MiFnYsk-QCMp1Zy3Xzw/project-details/10580096">https://reporter.nih.gov/search/qr4MiFnYsk-QCMp1Zy3Xzw/project-details/10580096</a>. Accessed February 23, 2023.
- 18. Sekhon M, Cartwright M, Francis JJ. Acceptability of healthcare interventions: an overview of reviews and development of a theoretical framework. *BMC Health Services Research*. 2017/01/26 2017;17(1):88.
- 19. Ortblad KF, Sekhon M, Wang L, et al. Acceptability Assessment in HIV Prevention and Treatment Intervention and Service Delivery Research: A Systematic Review and Qualitative Analysis. *AIDS Behav.* Jul 23 2022.
- 20. Doggett EG, Lanham M, Wilcher R, Gafos M, Karim QA, Heise L. Optimizing HIV prevention for women: a review of evidence from microbicide studies and considerations for gender-sensitive microbicide introduction. *J Int AIDS Soc.* 2015;18(1):20536.
- 21. Denzin NK, Lincoln YS. *Handbook of qualitative research*. 2nd ed. Thousand Oaks, Calif.: Sage Publications; 2000.
- 22. Miles MB, Huberman AM. *Qualitative data analysis: An expanded sourcebook, 2nd ed.* Thousand Oaks, CA, US: Sage Publications, Inc; 1994.
- 23. Macqueen K, McLellan-Lemal E, Bartholow K, Milstein B. Team-based codebook development: Structure, process, and agreement. *Handbook for Team-Based Qualitative Research*. 01/01 2008:119-135.
- 24. Hughes R. Considering the Vignette Technique and its Application to a Study of Drug Injecting and HIV Risk and Safer Behaviour. *Sociology of Health & Illness.* 1998;20(3):381-400.